CLINICAL TRIAL: NCT03903822
Title: A PHASE 2B, RANDOMIZED, DOUBLE BLIND, VEHICLE CONTROLLED, PARALLEL GROUP, DOSE RANGING STUDY TO ASSESS THE EFFICACY, SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-06700841 CREAM APPLIED ONCE OR TWICE DAILY FOR 6 WEEKS IN PARTICIPANTS WITH MILD OR MODERATE ATOPIC DERMATITIS
Brief Title: Dose Ranging Study to Assess Efficacy, Safety, Tolerability and Pharmacokinetics of PF-06700841 Topical Cream in Participants With Mild or Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7931022; 2018-003050-24 (EudraCT Number)
Record Dates: First submitted 2019-03-20; First posted 2019-04-04 (Actual); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis
Keywords: Mild-to-Moderate Atopic Dermatitis; topical
MeSH Terms: conditions — Dermatitis, Atopic | interventions — PF-06700841

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- PF-06700841 0.1% cream QD (Experimental): PF-06700841 0.1% cream applied once daily (QD)
  Interventions: Drug: PF-06700841
- PF-06700841 0.3% cream QD (Experimental): PF-06700841 0.3% cream applied once daily (QD)
  Interventions: Drug: PF-06700841
- PF-06700841 1% cream QD (Experimental): PF-06700841 1% cream applied once daily (QD)
  Interventions: Drug: PF-06700841
- PF-06700841 3% cream QD (Experimental): PF-06700841 3% cream applied once daily (QD)
  Interventions: Drug: PF-06700841
- PF-06700841 0.3% cream BID (Experimental): PF-06700841 0.3% cream applied twice daily (BID)
  Interventions: Drug: PF-06700841
- PF-06700841 1% cream BID (Experimental): PF-06700841 1% cream applied twice daily (BID)
  Interventions: Drug: PF-06700841
- Vehicle cream QD (Placebo Comparator): Vehicle cream applied once daily (QD)
  Interventions: Drug: Vehicle (Placebo)
- Vehicle cream BID (Placebo Comparator): Vehicle cream applied twice daily (BID)
  Interventions: Drug: Vehicle (Placebo)

INTERVENTIONS:
Drug: PF-06700841 — PF-06700841 topical cream
  Arms: PF-06700841 0.1% cream QD; PF-06700841 0.3% cream BID; PF-06700841 0.3% cream QD; PF-06700841 1% cream BID; PF-06700841 1% cream QD; PF-06700841 3% cream QD
Drug: Vehicle (Placebo) — Vehicle topical cream
  Arms: Vehicle cream BID; Vehicle cream QD

SUMMARY:
This study is being conducted to provide data on efficacy, safety, tolerability and PK of multiple topical formulation concentrations of PF-06700841 topical cream in the treatment of mild to moderate atopic dermatitis (AD). The study is intended to enable selection of the dose and dosing regimen (once daily [QD] vs twice daily [BID] application) for the future clinical development of topical PF-06700841.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Atopic Dermatitis for at least 3 months
* Investigator's Global Assessment (IGA) Score of 2 or 3
* Eczema Area Severity Index (EASI) score of 3-21
* Body Surface Area (BSA) of 2-20%
* Peak pruritus-Numerical Rating Scale (PPNRS) of Grade 2 or more

Exclusion Criteria:

* Other forms of dermatological diseases (other than atopic dermatitis)
* Fitzpatrick skin type score greater than 5
* Clinically significant abnormal ECG, vital signs, and laboratory values
* Infection with HBV, HCV, herpes zoster or tuberculosis

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (76):
- United States (36):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Center for Dermatology and Plastic Surgery/CCT, Scottsdale, Arizona
  - Center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - Beach Allergy and Asthma Specialty Group, A Medical Corporation, Long Beach, California
  - Clinical Science Institute, Santa Monica, California
  - New England Associates, LLC, Bridgeport, Connecticut
  - Dermatology Physicians of Connecticut, Shelton, Connecticut
  - Yolanda C. Holmes, MD, Washington D.C., District of Columbia
  - Olympian Clinical Research, Clearwater, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Precision Imaging, Jacksonville, Florida
  - Solutions Through Advanced Research, Inc, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Ormond Beach, Florida
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - DS Research, New Albany, Indiana
  - DS Research, Louisville, Kentucky
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Health Concepts, Rapid City, South Dakota
  - Tanenbaum Dermatology Center, Memphis, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - studies in Dermatology, LLC, Cypress, Texas
  - Center for Clinical Studies, LTD.LLP, Houston, Texas
  - Ventavia Research Group LLC, Hurst, Texas
  - Center for Clinical Studies, LTD. LLP, Webster, Texas
  - Summit Clinical Research, LLC, Franklin, Virginia
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
- Australia (4):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Emeritus Research, Camberwell, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Cabrini Hospital, Malvern, Victoria
- Bulgaria (3):
  - Center for Skin and Venereal Diseases EOOD - Sofia, Sofia
  - DCC Alexandrovska, Sofia
  - Diagnostic Consultative Center - Fokus-5 - Medical Establishment for Outpatient Care OOD, Sofia
- Canada (4):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SKiN Health, Cobourg, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Gentofte Hospital, Hellerup, Denmark
- Germany (10):
  - Emovis GmbH, Berlin
  - Rothhaar Studien GmbH, Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Klinikum Bielefeld gem.GmbH, Bielefeld
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Frankfurt, Frankfurt
  - MENSINGDERMA research GmbH, Hamburg
  - MVZ Alstermed GmbH, Hamburg
  - Dermatologische Gemeinschaftspraxis, Mahlow
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hungary (5):
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bacs-Kiskun Megyei Korhaz Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Oktato Korhaza, Kecskemét
  - CRU Hungary Kft., Miskolc
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Japan (6):
  - Kitago Dermatology Clinic, Sapporo, Hokkaido
  - Nakatsuhifuka Clinic, Kita-ku, Osaka-shi, Osaka
  - Parkside Hiroo Ladies Clinic, Minato-ku, Tokyo
  - Tanpopo Skin Clinic, Ōta-ku, Tokyo
  - Shinjuku Minamiguchi Dermatology Skin Clinic, Shinjuku-ku, Tokyo
  - Medical Corporation Jitai-kai Tachikawa Dermatology Clinic, Tachikawa, Tokyo
- Latvia (3):
  - Aesthetic dermatology clinic of Prof. J. Kisis, Riga
  - Health and Aesthetics Ltd, Riga
  - Outpatient Clinic of Ventspils, Ventspils
- Poland (4):
  - NZOZ Specjalistyczny Ośrodek Dermatologiczny DERMAL s.c., Bialystok
  - NASZ LEKARZ Przychodnie Medyczne, Torun
  - MTZ Clinical Research Sp. z o.o, Warsaw
  - WroMedica I. Bielicka, A. Strzalkowska s.c., Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931022

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Cream Once Daily (QD): Participants or caregivers of participants, topically applied vehicle cream on all eligible atopic dermatitis (AD) areas (of participants) once daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- PF-06700841 0.1% Cream QD: Participants or caregivers of participants, topically applied PF-06700841 0.1 percent (%) cream on all eligible AD areas (of participants) once daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- PF-06700841 0.3% Cream QD: Participants or caregivers of participants, topically applied PF-06700841 0.3 % cream on all eligible AD areas (of participants) once daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- PF-06700841 1.0% Cream QD: Participants or caregivers of participants, topically applied PF-06700841 1.0 % cream on all eligible AD areas (of participants) once daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- PF-06700841 3.0% Cream QD: Participants or caregivers of participants, topically applied PF-06700841 3.0 % cream on all eligible AD areas (of participants) once daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- Vehicle Cream Twice Daily (BID): Participants or caregivers of participants, topically applied vehicle cream on all eligible AD areas (of participants) twice daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- PF-06700841 0.3% Cream BID: Participants or caregivers of participants, topically applied PF-06700841 0.3% cream on all eligible AD areas (of participants) twice daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- PF-06700841 1.0% Cream BID: Participants or caregivers of participants, topically applied PF-06700841 1.0 % cream on all eligible AD areas (of participants) twice daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
Period: Treatment Phase (6 Weeks)
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Started | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Completed | 28 | 27 | 33 | 32 | 31 | 25 | 31 | 33
Not Completed | 9 | 10 | 3 | 5 | 5 | 11 | 5 | 4
Not completed — Adverse Event | 3 | 3 | 1 | 1 | 1 | 6 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 2 | 2 | 1 | 2 | 3 | 3
Not completed — Refused Further Treatment | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Period: Follow up Phase (4 Weeks)
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Started | 37 (Participants not completing treatment phase could also start this phase.) | 37 (Participants not completing treatment phase could also start this phase.) | 36 (Participants not completing treatment phase could also start this phase.) | 37 (Participants not completing treatment phase could also start this phase.) | 36 (Participants not completing treatment phase could also start this phase.) | 36 (Participants not completing treatment phase could also start this phase.) | 36 (Participants not completing treatment phase could also start this phase.) | 37 (Participants not completing treatment phase could also start this phase.)
Completed | 29 | 29 | 32 | 33 | 32 | 28 | 31 | 31
Not Completed | 8 | 8 | 4 | 4 | 4 | 8 | 5 | 6
Not completed — Adverse Event | 3 | 2 | 1 | 1 | 0 | 5 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 3 | 2 | 2 | 2 | 3 | 3
Not completed — Refused Further Study Procedures | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug.
Groups:
- Vehicle Cream Once Daily (QD): Participants or caregivers of participants, topically applied vehicle cream on all eligible AD areas (of participants) once daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- PF-06700841 0.1% Cream QD: Participants or caregivers of participants, topically applied PF-06700841 0.1 % cream on all eligible AD areas (of participants) once daily for a maximum of 6 weeks. Eligibility of AD areas to be treated were determined on Day 1 by investigator. Participants were followed up for 4 weeks after last dose.
- Total: Total of all reporting groups
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID | Total
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37 | 292
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (16.80) | 40.8 (15.35) | 43.4 (16.43) | 38.4 (12.90) | 40.5 (12.30) | 42.3 (18.18) | 39.4 (17.27) | 38.1 (15.34) | 40.2 (15.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 24 | 23 | 15 | 19 | 16 | 20 | 156
  Male | 17 | 18 | 12 | 14 | 21 | 17 | 20 | 17 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 2 | 1 | 3 | 0 | 4 | 13
  Not Hispanic or Latino | 37 | 37 | 32 | 35 | 35 | 33 | 35 | 33 | 277
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 8 | 4 | 8 | 10 | 9 | 9 | 7 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Black or African American | 8 | 7 | 9 | 6 | 4 | 6 | 5 | 6 | 51
  White | 24 | 22 | 21 | 20 | 21 | 20 | 22 | 24 | 174
  More than one race | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 5
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 6: Multiple Imputation
Description: EASI evaluates severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions(head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in each 4 body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Week 6
Population: Full analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug. Missing data were imputed with multiple imputation method assuming responses are similar to the corresponding vehicle arm under the MAR assumption
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Percent change | -44.4 [-57.3 to -31.6] | -58.3 [-71.2 to -45.5] | -64.6 [-77.1 to -52.1] | -70.1 [-82.1 to -58.0] | -67.9 [-80.6 to -55.3] | -47.6 [-57.5 to -37.7] | -58.6 [-67.5 to -49.7] | -75.0 [-83.8 to -66.2]
Statistical Analysis 1: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; Analysis of covariance (ANCOVA) contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.1040, ANCOVA; Least square (LS) mean difference = -13.9, 90% CI 2-sided [-32.1 to 4.3], Standard Error of Mean 11.04
Statistical Analysis 2: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0334, ANCOVA; LS Mean Difference = -20.2, 90% CI 2-sided [-38.3 to -2.1], Standard Error of Mean 11.00
Statistical Analysis 3: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0086, ANCOVA; LS Mean Difference = -25.6, 90% CI 2-sided [-43.3 to -8.0], Standard Error of Mean 10.75
Statistical Analysis 4: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0158, ANCOVA; LS Mean Difference = -23.5, 90% CI 2-sided [-41.5 to -5.5], Standard Error of Mean 10.93
Statistical Analysis 5: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0879, ANCOVA; LS Mean Difference = -11.0, 90% CI 2-sided [-24.3 to 2.4], Standard Error of Mean 8.11
Statistical Analysis 6: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -27.4, 90% CI 2-sided [-40.7 to -14.1], Standard Error of Mean 8.11

2. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Score Clear (0) or Almost Clear (1) and a Reduction From Baseline of Greater Than or Equal to ( >=2) Points at Week 6: Non-responder Imputation
Description: IGA assesses severity of participant's AD on a 5 point scale. 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting and 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Higher scores indicating more severity of AD. Assessment excluded soles, palms and scalp.
Time Frame: Baseline, Week 6
Population: Full analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug. Non-Responder Imputation (NRI) method: participants with missing values were considered to be non-responders.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Percentage of participants | 10.8 [4.8 to 22.2] | 29.7 [18.5 to 43.3] | 33.3 [21.3 to 47.0] | 40.5 [28.0 to 54.4] | 44.4 [30.2 to 59.1] | 13.9 [6.9 to 25.4] | 33.3 [21.3 to 47.0] | 27.0 [15.5 to 40.2]
Statistical Analysis 1: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0244, Chan and Zhang Exact Method; Risk Difference (RD) = 18.9, 90% CI 2-sided [2.4 to 34.7]
Statistical Analysis 2: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0113, Chan and Zhang Exact Method; Risk Difference (RD) = 22.5, 90% CI 2-sided [4.8 to 38.6]
Statistical Analysis 3: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0018, Chan and Zhang Exact Method; Risk Difference (RD) = 29.7, 90% CI 2-sided [11.0 to 45.7]
Statistical Analysis 4: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0007, Chan and Zhang Exact Method; Risk Difference (RD) = 33.6, 90% CI 2-sided [13.7 to 49.9]
Statistical Analysis 5: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0289, Chan and Zhang Exact Method; Risk Difference (RD) = 19.4, 90% CI 2-sided [1.8 to 36.5]
Statistical Analysis 6: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1145, Chan and Zhang Exact Method; Risk Difference (RD) = 13.1, 90% CI 2-sided [-2.9 to 29.6]

3. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 6: Multiple Imputation
Description: as for outcome 1
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Units on a scale | -3.2 [-4.1 to -2.3] | -4.5 [-5.4 to -3.6] | -4.6 [-5.5 to -3.7] | -4.8 [-5.7 to -3.9] | -5.5 [-6.4 to -4.7] | -3.6 [-4.3 to -3.0] | -4.4 [-5.0 to -3.8] | -5.3 [-5.9 to -4.7]
Statistical Analysis 1: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0488, ANCOVA; LS mean difference = -1.31, 90% CI 2-sided [-2.61 to -0.01], Standard Error of Mean 0.790
Statistical Analysis 2: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0413, ANCOVA; LS Mean Difference = -1.37, 90% CI 2-sided [-2.66 to -0.07], Standard Error of Mean 0.788
Statistical Analysis 3: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0200, ANCOVA; LS Mean Difference = -1.59, 90% CI 2-sided [-2.86 to -0.32], Standard Error of Mean 0.773
Statistical Analysis 4: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0011, ANCOVA; LS Mean Difference = -2.33, 90% CI 2-sided [-3.58 to -1.08], Standard Error of Mean 0.758
Statistical Analysis 5: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0727, ANCOVA; LS Mean Difference = -0.78, 90% CI 2-sided [-1.66 to 0.10], Standard Error of Mean 0.535
Statistical Analysis 6: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; ANCOVA contained fixed factors of treatment and baseline value; Test type: Superiority; p = 0.0010, ANCOVA; LS Mean Difference = -1.64, 90% CI 2-sided [-2.52 to -0.77], Standard Error of Mean 0.534

4. Secondary Outcome: Percentage of Participants Achieving >=2 Points Reduction in Peak Pruritus Numerical Rating Scale (PP-NRS) From Baseline at Weeks 1, 2, 3, 4 and 6: Non-responder Imputation
Description: The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants at specified time points were asked the following question: "How would you rate your itch due to AD at the worst moment during the previous 24 hours?" The scale ranged from 0-10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Time Frame: Baseline, Weeks 1, 2, 3, 4 and 6
Population: Full analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. NRI method: participants with missing values were considered to be non-responders.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 36 | 35 | 37 | 36 | 36 | 35 | 35
Percentage of participants
  At Week 1 | 16.2 [7.3 to 29.3] | 16.7 [7.5 to 30.2] | 20.0 [11.0 to 33.8] | 29.7 [18.5 to 43.3] | 44.4 [30.2 to 59.1] | 13.9 [6.9 to 25.4] | 28.6 [16.4 to 41.9] | 25.7 [15.4 to 39.2]
  At Week 2 | 24.3 [14.5 to 37.0] | 30.6 [18.9 to 44.0] | 42.9 [30.0 to 58.1] | 48.6 [34.3 to 63.0] | 61.1 [47.0 to 74.6] | 25.0 [14.9 to 38.0] | 45.7 [31.7 to 60.8] | 37.1 [23.6 to 52.2]
  At Week 3 | 21.6 [11.2 to 34.3] | 38.9 [25.4 to 53.0] | 48.6 [33.8 to 63.5] | 59.5 [45.6 to 72.0] | 58.3 [44.0 to 71.0] | 33.3 [21.3 to 47.0] | 51.4 [36.5 to 66.2] | 57.1 [41.9 to 70.0]
  At Week 4 | 35.1 [22.2 to 49.3] | 38.9 [25.4 to 53.0] | 51.4 [36.5 to 66.2] | 62.2 [48.0 to 75.2] | 58.3 [44.0 to 71.0] | 30.6 [18.9 to 44.0] | 60.0 [44.8 to 74.0] | 60.0 [44.8 to 74.0]
  At Week 6 | 40.5 [28.0 to 54.4] | 41.7 [29.0 to 56.0] | 51.4 [36.5 to 66.2] | 56.8 [43.2 to 70.7] | 61.1 [47.0 to 74.6] | 30.6 [18.9 to 44.0] | 60.0 [44.8 to 74.0] | 60.0 [44.8 to 74.0]
Statistical Analysis 1: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.5246, Chan and Zhang Exact Method; Risk Difference (RD) = 0.5, 90% CI 2-sided [-14.7 to 16.4]
Statistical Analysis 2: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.3906, Chan and Zhang Exact Method; Risk Difference (RD) = 3.8, 90% CI 2-sided [-12.5 to 19.9]
Statistical Analysis 3: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1193, Chan and Zhang Exact Method; Risk Difference (RD) = 13.5, 90% CI 2-sided [-3.2 to 30.6]
Statistical Analysis 4: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0048, Chan and Zhang Exact Method; Risk Difference (RD) = 28.2, 90% CI 2-sided [8.8 to 45.5]
Statistical Analysis 5: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0777, Chan and Zhang Exact Method; Risk Difference (RD) = 14.7, 90% CI 2-sided [-2.0 to 31.1]
Statistical Analysis 6: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1245, Chan and Zhang Exact Method; Risk Difference (RD) = 11.8, 90% CI 2-sided [-4.3 to 28.0]
Statistical Analysis 7: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.3322, Chan and Zhang Exact Method; Risk Difference (RD) = 6.2, 90% CI 2-sided [-12.2 to 24.4]
Statistical Analysis 8: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0535, Chan and Zhang Exact Method; Risk Difference (RD) = 18.5, 90% CI 2-sided [-0.3 to 36.5]
Statistical Analysis 9: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0159, Chan and Zhang Exact Method; Risk Difference (RD) = 24.3, 90% CI 2-sided [4.5 to 41.9]
Statistical Analysis 10: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0008, Chan and Zhang Exact Method; Risk Difference (RD) = 36.8, 90% CI 2-sided [15.4 to 54.0]
Statistical Analysis 11: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0386, Chan and Zhang Exact Method; Risk Difference (RD) = 20.7, 90% CI 2-sided [1.5 to 38.8]
Statistical Analysis 12: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1485, Chan and Zhang Exact Method; Risk Difference (RD) = 12.1, 90% CI 2-sided [-6.4 to 30.3]
Statistical Analysis 13: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0620, Chan and Zhang Exact Method; Risk Difference (RD) = 17.3, 90% CI 2-sided [-0.8 to 34.8]
Statistical Analysis 14: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0089, Chan and Zhang Exact Method; Risk Difference (RD) = 26.9, 90% CI 2-sided [6.5 to 44.4]
Statistical Analysis 15: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0005, Chan and Zhang Exact Method; Risk Difference (RD) = 37.8, 90% CI 2-sided [17.5 to 54.7]
Statistical Analysis 16: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0007, Chan and Zhang Exact Method; Risk Difference (RD) = 36.7, 90% CI 2-sided [15.4 to 54.0]
Statistical Analysis 17: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0711, Chan and Zhang Exact Method; Risk Difference (RD) = 18.1, 90% CI 2-sided [-2.0 to 37.5]
Statistical Analysis 18: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0266, Chan and Zhang Exact Method; Risk Difference (RD) = 23.8, 90% CI 2-sided [2.7 to 42.5]
Statistical Analysis 19: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.4173, Chan and Zhang Exact Method; Risk Difference (RD) = 3.8, 90% CI 2-sided [-15.3 to 23.1]
Statistical Analysis 20: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1096, Chan and Zhang Exact Method; Risk Difference (RD) = 16.3, 90% CI 2-sided [-4.3 to 35.6]
Statistical Analysis 21: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0133, Chan and Zhang Exact Method; Risk Difference (RD) = 27.0, 90% CI 2-sided [6.1 to 45.7]
Statistical Analysis 22: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0304, Chan and Zhang Exact Method; Risk Difference (RD) = 23.2, 90% CI 2-sided [2.6 to 41.7]
Statistical Analysis 23: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0078, Chan and Zhang Exact Method; Risk Difference (RD) = 29.4, 90% CI 2-sided [7.2 to 47.6]
Statistical Analysis 24: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0078, Chan and Zhang Exact Method; Risk Difference (RD) = 29.4, 90% CI 2-sided [7.2 to 47.6]
Statistical Analysis 25: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.4966, Chan and Zhang Exact Method; Risk Difference (RD) = 1.1, 90% CI 2-sided [-18.4 to 20.4]
Statistical Analysis 26: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.2753, Chan and Zhang Exact Method; Risk Difference (RD) = 10.9, 90% CI 2-sided [-9.3 to 30.1]
Statistical Analysis 27: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1036, Chan and Zhang Exact Method; Risk Difference (RD) = 16.2, 90% CI 2-sided [-4.2 to 35.7]
Statistical Analysis 28: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0457, Chan and Zhang Exact Method; Risk Difference (RD) = 20.6, 90% CI 2-sided [0.4 to 39.6]
Statistical Analysis 29: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0078, Chan and Zhang Exact Method; Risk Difference (RD) = 29.4, 90% CI 2-sided [7.2 to 47.6]
Statistical Analysis 30: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0078, Chan and Zhang Exact Method; Risk Difference (RD) = 29.4, 90% CI 2-sided [7.2 to 47.6]

5. Secondary Outcome: Percentage of Participants Achieving >=4 Points Reduction in Peak Pruritus Numerical Rating Scale (PP-NRS) From Baseline at Weeks 1, 2, 3, 4, 6 and Follow-up Visit: Non-responder Imputation
Description: as for outcome 4
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 33 | 30 | 32 | 31 | 28 | 30 | 30 | 27
Percentage of participants
  At Week 1 | 0.0 [0.0 to 8.2] | 3.3 [0.4 to 14.0] | 3.1 [0.3 to 13.1] | 16.1 [8.1 to 29.7] | 10.7 [4.0 to 23.8] | 3.3 [0.4 to 14.0] | 3.3 [0.4 to 14.0] | 11.1 [4.2 to 24.8]
  At Week 2 | 9.1 [3.4 to 20.2] | 10.0 [3.7 to 22.1] | 9.4 [3.5 to 20.7] | 19.4 [8.8 to 32.7] | 25.0 [13.9 to 40.0] | 10.0 [3.7 to 22.1] | 13.3 [5.9 to 27.9] | 33.3 [20.4 to 50.0]
  At Week 3 | 12.1 [5.4 to 25.1] | 23.3 [12.9 to 37.6] | 15.6 [7.8 to 28.7] | 32.3 [18.7 to 48.2] | 32.1 [19.7 to 47.3] | 10.0 [3.7 to 22.1] | 20.0 [9.1 to 33.9] | 37.0 [22.1 to 54.7]
  At Week 4 | 18.2 [8.2 to 31.3] | 26.7 [14.0 to 41.6] | 28.1 [17.0 to 43.3] | 35.5 [21.3 to 51.8] | 50.0 [33.3 to 66.7] | 10.0 [3.7 to 22.1] | 30.0 [18.2 to 45.5] | 37.0 [22.1 to 54.7]
  At Week 6 | 18.2 [8.2 to 31.3] | 30.0 [18.2 to 45.5] | 34.4 [20.7 to 50.0] | 45.2 [29.7 to 60.1] | 50.0 [33.3 to 66.7] | 16.7 [8.3 to 30.8] | 33.3 [19.3 to 49.2] | 40.7 [24.8 to 58.3]
  At Follow-up visit | 9.1 [3.4 to 20.2] | 30.0 [18.2 to 45.5] | 21.9 [12.1 to 36.2] | 19.4 [8.8 to 32.7] | 21.4 [9.8 to 36.6] | 20.0 [9.1 to 33.9] | 20.0 [9.1 to 33.9] | 7.4 [2.0 to 20.4]
Statistical Analysis 1: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.2450, Chan and Zhang Exact Method; Risk Difference (RD) = 3.3, 90% CI 2-sided [-5.4 to 14.9]
Statistical Analysis 2: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.2575, Chan and Zhang Exact Method; Risk Difference (RD) = 3.1, 90% CI 2-sided [-5.3 to 14.0]
Statistical Analysis 3: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0087, Chan and Zhang Exact Method; Risk Difference (RD) = 16.1, 90% CI 2-sided [5.7 to 31.0]
Statistical Analysis 4: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0392, Chan and Zhang Exact Method; Risk Difference (RD) = 10.7, 90% CI 2-sided [0.8 to 25.4]
Statistical Analysis 5: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 1.0000, Chan and Zhang Exact Method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-11.2 to 11.2]
Statistical Analysis 6: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1528, Chan and Zhang Exact Method; Risk Difference (RD) = 7.8, 90% CI 2-sided [-4.9 to 22.5]
Statistical Analysis 7: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.4989, Chan and Zhang Exact Method; Risk Difference (RD) = 0.9, 90% CI 2-sided [-12.7 to 15.2]
Statistical Analysis 8: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.5419, Chan and Zhang Exact Method; Risk Difference (RD) = 0.3, 90% CI 2-sided [-13.6 to 14.2]
Statistical Analysis 9: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1362, Chan and Zhang Exact Method; Risk Difference (RD) = 10.3, 90% CI 2-sided [-5.0 to 26.2]
Statistical Analysis 10: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0541, Chan and Zhang Exact Method; Risk Difference (RD) = 15.9, 90% CI 2-sided [-0.4 to 33.9]
Statistical Analysis 11: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.3945, Chan and Zhang Exact Method; Risk Difference (RD) = 3.3, 90% CI 2-sided [-12.0 to 19.5]
Statistical Analysis 12: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0201, Chan and Zhang Exact Method; Risk Difference (RD) = 23.3, 90% CI 2-sided [3.9 to 41.8]
Statistical Analysis 13: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1372, Chan and Zhang Exact Method; Risk Difference (RD) = 11.2, 90% CI 2-sided [-5.4 to 28.2]
Statistical Analysis 14: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.3924, Chan and Zhang Exact Method; Risk Difference (RD) = 3.5, 90% CI 2-sided [-11.6 to 19.1]
Statistical Analysis 15: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0311, Chan and Zhang Exact Method; Risk Difference (RD) = 20.1, 90% CI 2-sided [2.4 to 38.3]
Statistical Analysis 16: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0392, Chan and Zhang Exact Method; Risk Difference (RD) = 20.0, 90% CI 2-sided [0.8 to 38.1]
Statistical Analysis 17: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1541, Chan and Zhang Exact Method; Risk Difference (RD) = 10.0, 90% CI 2-sided [-6.2 to 26.4]
Statistical Analysis 18: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0091, Chan and Zhang Exact Method; Risk Difference (RD) = 27.0, 90% CI 2-sided [6.8 to 45.4]
Statistical Analysis 19: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.2835, Chan and Zhang Exact Method; Risk Difference (RD) = 8.5, 90% CI 2-sided [-9.5 to 27.0]
Statistical Analysis 20: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.2700, Chan and Zhang Exact Method; Risk Difference (RD) = 9.9, 90% CI 2-sided [-8.7 to 27.8]
Statistical Analysis 21: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0662, Chan and Zhang Exact Method; Risk Difference (RD) = 17.3, 90% CI 2-sided [-1.4 to 36.2]
Statistical Analysis 22: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0050, Chan and Zhang Exact Method; Risk Difference (RD) = 31.8, 90% CI 2-sided [9.2 to 50.4]
Statistical Analysis 23: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0302, Chan and Zhang Exact Method; Risk Difference (RD) = 20.0, 90% CI 2-sided [2.2 to 38.3]
Statistical Analysis 24: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0091, Chan and Zhang Exact Method; Risk Difference (RD) = 27.0, 90% CI 2-sided [6.8 to 45.4]
Statistical Analysis 25: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1561, Chan and Zhang Exact Method; Risk Difference (RD) = 11.8, 90% CI 2-sided [-6.5 to 30.2]
Statistical Analysis 26: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0753, Chan and Zhang Exact Method; Risk Difference (RD) = 16.2, 90% CI 2-sided [-2.7 to 34.8]
Statistical Analysis 27: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0108, Chan and Zhang Exact Method; Risk Difference (RD) = 27.0, 90% CI 2-sided [5.7 to 46.0]
Statistical Analysis 28: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0050, Chan and Zhang Exact Method; Risk Difference (RD) = 31.8, 90% CI 2-sided [9.2 to 50.4]
Statistical Analysis 29: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0775, Chan and Zhang Exact Method; Risk Difference (RD) = 16.7, 90% CI 2-sided [-2.9 to 35.7]
Statistical Analysis 30: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0243, Chan and Zhang Exact Method; Risk Difference (RD) = 24.1, 90% CI 2-sided [3.4 to 43.4]
Statistical Analysis 31: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At follow-up visit: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0234, Chan and Zhang Exact Method; Risk Difference (RD) = 20.9, 90% CI 2-sided [3.5 to 38.8]
Statistical Analysis 32: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At follow-up visit: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1134, Chan and Zhang Exact Method; Risk Difference (RD) = 12.8, 90% CI 2-sided [-2.8 to 29.3]
Statistical Analysis 33: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At follow-up visit: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1362, Chan and Zhang Exact Method; Risk Difference (RD) = 10.3, 90% CI 2-sided [-5.0 to 26.2]
Statistical Analysis 34: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At follow-up visit: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1029, Chan and Zhang Exact Method; Risk Difference (RD) = 12.3, 90% CI 2-sided [-3.4 to 29.8]
Statistical Analysis 35: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At follow-up visit: Risk difference = difference in percentage of participants; Test type: Superiority; p = 1.0000, Chan and Zhang Exact Method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-17.9 to 17.9]
Statistical Analysis 36: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At follow-up visit: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.8972, Chan and Zhang Exact Method; Risk Difference (RD) = -12.6, 90% CI 2-sided [-28.8 to 3.5]

6. Secondary Outcome: Percent Change From Baseline in Affected Body Surface Area (BSA) at Weeks 1, 2, 3, 4, 6 and Follow-up Visit
Description: 4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: Full analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the each specified time point.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 34 | 36 | 33 | 35 | 34 | 34 | 36 | 36
Percent change
  At Week 1 | -2.4 [-12.2 to 7.4] | -2.9 [-12.5 to 6.8] | -16.2 [-26.2 to -6.2] | -19.9 [-29.6 to -10.2] | -23.0 [-32.8 to -13.1] | 8.5 [-8.3 to 25.3] | -16.5 [-32.9 to -0.1] | -17.0 [-33.5 to -0.5]
  At Week 2: number analyzed (Participants) | 34 | 33 | 33 | 33 | 32 | 32 | 33 | 32
  At Week 2 | -15.3 [-28.0 to -2.6] | -7.2 [-20.2 to 5.8] | -38.1 [-51.0 to -25.2] | -43.6 [-56.5 to -30.8] | -39.0 [-52.1 to -26.0] | -2.5 [-14.0 to 9.1] | -34.2 [-45.4 to -22.9] | -43.1 [-54.5 to -31.6]
  At Week 3: number analyzed (Participants) | 28 | 29 | 32 | 34 | 31 | 23 | 30 | 33
  At Week 3 | -17.1 [-31.0 to -3.1] | -13.1 [-27.4 to 1.1] | -50.6 [-64.4 to -36.7] | -55.9 [-69.7 to -42.0] | -49.2 [-63.2 to -35.1] | -25.2 [-39.2 to -11.1] | -39.8 [-53.0 to -26.6] | -44.0 [-57.1 to -30.9]
  At Week 4: number analyzed (Participants) | 30 | 28 | 33 | 32 | 32 | 25 | 32 | 32
  At Week 4 | -25.9 [-39.8 to -12.0] | -20.1 [-34.4 to -5.7] | -55.8 [-69.5 to -42.1] | -57.9 [-71.7 to -44.0] | -56.7 [-70.8 to -42.7] | -34.7 [-46.1 to -23.3] | -46.4 [-56.9 to -35.9] | -57.7 [-68.2 to -47.2]
  At Week 6: number analyzed (Participants) | 29 | 28 | 31 | 32 | 31 | 24 | 32 | 33
  At Week 6 | -21.6 [-38.0 to -5.3] | -39.4 [-56.1 to -22.7] | -59.4 [-75.4 to -43.5] | -63.6 [-79.5 to -47.6] | -60.3 [-76.4 to -44.1] | -31.2 [-42.5 to -20.0] | -48.9 [-59.3 to -38.6] | -65.0 [-75.3 to -54.7]
  At Follow-up visit: number analyzed (Participants) | 29 | 27 | 32 | 31 | 26 | 28 | 30 | 29
  At Follow-up visit | -23.6 [-39.5 to -7.6] | -24.5 [-41.0 to -8.0] | -42.7 [-58.1 to -27.2] | -37.0 [-52.6 to -21.4] | -55.2 [-71.8 to -38.6] | -26.3 [-47.5 to -5.2] | -31.6 [-52.0 to -11.3] | -24.6 [-45.2 to -4.1]
Statistical Analysis 1: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 1: Mixed Model Repeated Measure (MMRM) contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.4781, Mixed Model Repeated Measure; LS Mean difference = -0.5, 90% CI 2-sided [-14.2 to 13.3], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 1: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0522, Mixed Model Repeated Measure; LS Mean difference = -13.8, 90% CI 2-sided [-27.8 to 0.2], Standard Error of Mean 8.47
Statistical Analysis 3: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 1: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0187, Mixed Model Repeated Measure; LS Mean difference = -17.5, 90% CI 2-sided [-31.4 to -3.7], Standard Error of Mean 8.37
Statistical Analysis 4: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 1: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0080, Mixed Model Repeated Measure; LS Mean difference = -20.6, 90% CI 2-sided [-34.5 to -6.6], Standard Error of Mean 8.45
Statistical Analysis 5: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 1: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0401, Mixed Model Repeated Measure; LS Mean difference = -25.0, 90% CI 2-sided [-48.6 to -1.5], Standard Error of Mean 14.17
Statistical Analysis 6: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 1: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0379, Mixed Model Repeated Measure; LS Mean difference = -25.5, 90% CI 2-sided [-49.2 to -1.9], Standard Error of Mean 14.25
Statistical Analysis 7: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 2: MMRM contained fixed factors of treatment, visit(Weeks 1, 2, 3, 4, 6 and follow up), treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.7678, Mixed Model Repeated Measure; LS Mean difference = 8.1, 90% CI 2-sided [-10.1 to 26.3], Standard Error of Mean 11.01
Statistical Analysis 8: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 2: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0193, Mixed Model Repeated Measure; LS Mean difference = -22.8, 90% CI 2-sided [-40.9 to -4.7], Standard Error of Mean 10.94
Statistical Analysis 9: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 2:MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0052, Mixed Model Repeated Measure; LS Mean difference = -28.3, 90% CI 2-sided [-46.5 to -10.2], Standard Error of Mean 10.95
Statistical Analysis 10: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 2: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0164, Mixed Model Repeated Measure; LS Mean difference = -23.7, 90% CI 2-sided [-42.0 to -5.5], Standard Error of Mean 11.03
Statistical Analysis 11: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 2: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0008, Mixed Model Repeated Measure; LS Mean difference = -31.7, 90% CI 2-sided [-47.8 to -15.6], Standard Error of Mean 9.72
Statistical Analysis 12: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 2: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p < 0.0001, Mixed Model Repeated Measure; LS Mean difference = -40.6, 90% CI 2-sided [-57.0 to -24.3], Standard Error of Mean 9.86
Statistical Analysis 13: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 3: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.6269, Mixed Model Repeated Measure; LS Mean difference = 3.9, 90% CI 2-sided [-16.1 to 23.9], Standard Error of Mean 12.09
Statistical Analysis 14: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 3: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0027, Mixed Model Repeated Measure; LS Mean difference = -33.5, 90% CI 2-sided [-53.1 to -13.8], Standard Error of Mean 11.87
Statistical Analysis 15: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 3: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0007, Mixed Model Repeated Measure; LS Mean difference = -38.8, 90% CI 2-sided [-58.5 to -19.2], Standard Error of Mean 11.89
Statistical Analysis 16: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 3: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0041, Mixed Model Repeated Measure; LS Mean difference = -32.1, 90% CI 2-sided [-51.9 to -12.3], Standard Error of Mean 12.00
Statistical Analysis 17: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 3: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.1054, Mixed Model Repeated Measure; LS Mean difference = -14.6, 90% CI 2-sided [-33.9 to 4.6], Standard Error of Mean 11.61
Statistical Analysis 18: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 3: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0542, Mixed Model Repeated Measure; LS Mean difference = -18.8, 90% CI 2-sided [-38.1 to 0.5], Standard Error of Mean 11.62
Statistical Analysis 19: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 4: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.6847, Mixed Model Repeated Measure; LS Mean difference = 5.8, 90% CI 2-sided [-14.2 to 25.9], Standard Error of Mean 12.12
Statistical Analysis 20: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 4: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0062, Mixed Model Repeated Measure; LS Mean difference = -29.9, 90% CI 2-sided [-49.4 to -10.3], Standard Error of Mean 11.82
Statistical Analysis 21: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 4: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0040, Mixed Model Repeated Measure; LS Mean difference = -32.0, 90% CI 2-sided [-51.6 to -12.3], Standard Error of Mean 11.89
Statistical Analysis 22: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 4: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0054, Mixed Model Repeated Measure; LS Mean difference = -30.8, 90% CI 2-sided [-50.6 to -11.0], Standard Error of Mean 11.97
Statistical Analysis 23: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 4: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.1076, Mixed Model Repeated Measure; LS Mean difference = -11.7, 90% CI 2-sided [-27.2 to 3.9], Standard Error of Mean 9.35
Statistical Analysis 24: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 4: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0082, Mixed Model Repeated Measure; LS Mean difference = -23.0, 90% CI 2-sided [-38.6 to -7.3], Standard Error of Mean 9.42
Statistical Analysis 25: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 6: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.1051, Mixed Model Repeated Measure; LS Mean difference = -17.8, 90% CI 2-sided [-41.2 to 5.6], Standard Error of Mean 14.14
Statistical Analysis 26: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 6: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0034, Mixed Model Repeated Measure; LS Mean difference = -37.8, 90% CI 2-sided [-60.6 to -15.0], Standard Error of Mean 13.80
Statistical Analysis 27: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 6: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0014, Mixed Model Repeated Measure; LS Mean difference = -41.9, 90% CI 2-sided [-64.8 to -19.0], Standard Error of Mean 13.83
Statistical Analysis 28: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 6: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0030, Mixed Model Repeated Measure; LS Mean difference = -38.6, 90% CI 2-sided [-61.6 to -15.6], Standard Error of Mean 13.90
Statistical Analysis 29: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 6: MMRM contained fixed factors of treatment, visit(Weeks 1, 2, 3, 4, 6 and follow up), treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0289, Mixed Model Repeated Measure; LS Mean difference = -17.7, 90% CI 2-sided [-33.0 to -2.4], Standard Error of Mean 9.22
Statistical Analysis 30: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 6: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0002, Mixed Model Repeated Measure; LS Mean difference = -33.8, 90% CI 2-sided [-49.2 to -18.4], Standard Error of Mean 9.27
Statistical Analysis 31: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At follow-up visit: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.4739, Mixed Model Repeated Measure; LS Mean difference = -0.9, 90% CI 2-sided [-23.9 to 22.0], Standard Error of Mean 13.88
Statistical Analysis 32: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At follow-up visit: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0789, Mixed Model Repeated Measure; LS Mean difference = -19.1, 90% CI 2-sided [-41.3 to 3.2], Standard Error of Mean 13.43
Statistical Analysis 33: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At follow-up visit: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.1611, Mixed Model Repeated Measure; LS Mean difference = -13.4, 90% CI 2-sided [-35.7 to 8.9], Standard Error of Mean 13.50
Statistical Analysis 34: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At follow-up visit: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.0124, Mixed Model Repeated Measure; LS Mean Difference = -31.6, 90% CI 2-sided [-54.7 to -8.5], Standard Error of Mean 13.94
Statistical Analysis 35: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At follow-up visit: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.3828, Mixed Model Repeated Measure; LS Mean difference = -5.3, 90% CI 2-sided [-34.7 to 24.1], Standard Error of Mean 17.68
Statistical Analysis 36: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At follow-up visit: MMRM contained fixed factors of treatment, visit, treatment-by-visit interaction and baseline value; Test type: Superiority; p = 0.5383, Mixed Model Repeated Measure; LS Mean difference = 1.7, 90% CI 2-sided [-27.9 to 31.3], Standard Error of Mean 17.80

7. Secondary Outcome: Percentage of Participants Achieving >=75% Improvement in Eczema Area and Severity Index Total Score (EASI-75) From Baseline at Weeks 1, 2, 3, 4 and 6: Non-responder Imputation
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 2, 3, 4 and 6
Population: Full analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug. NRI method: participants with missing values were considered to be non-responders.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Percentage of participants
  At Week 1 | 5.4 [1.4 to 15.5] | 0.0 [0.0 to 7.3] | 19.4 [10.7 to 32.8] | 5.4 [1.4 to 15.5] | 16.7 [7.5 to 30.2] | 0.0 [0.0 to 7.5] | 13.9 [6.9 to 25.4] | 21.6 [11.2 to 34.3]
  At Week 2 | 8.1 [3.0 to 18.5] | 10.8 [4.8 to 22.2] | 27.8 [15.9 to 40.9] | 24.3 [14.5 to 37.0] | 38.9 [25.4 to 53.0] | 13.9 [6.9 to 25.4] | 25.0 [14.9 to 38.0] | 32.4 [20.6 to 46.4]
  At Week 3 | 5.4 [1.4 to 15.5] | 16.2 [7.3 to 29.3] | 36.1 [22.9 to 50.0] | 43.2 [29.3 to 56.8] | 41.7 [29.0 to 56.0] | 19.4 [10.7 to 32.8] | 19.4 [10.7 to 32.8] | 43.2 [29.3 to 56.8]
  At Week 4 | 24.3 [14.5 to 37.0] | 21.6 [11.2 to 34.3] | 38.9 [25.4 to 53.0] | 43.2 [29.3 to 56.8] | 50.0 [35.3 to 64.7] | 22.2 [11.6 to 35.3] | 36.1 [22.9 to 50.0] | 48.6 [34.3 to 63.0]
  At Week 6 | 35.1 [22.2 to 49.3] | 32.4 [20.6 to 46.4] | 52.8 [38.0 to 67.2] | 54.1 [40.2 to 68.2] | 50.0 [35.3 to 64.7] | 16.7 [7.5 to 30.2] | 36.1 [22.9 to 50.0] | 51.4 [37.0 to 65.7]
Statistical Analysis 1: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.8964, Chan and Zhang Exact Method; Risk Difference (RD) = -5.4, 90% CI 2-sided [-16.1 to 2.0]
Statistical Analysis 2: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0391, Chan and Zhang Exact Method; Risk Difference (RD) = 14.0, 90% CI 2-sided [1.0 to 28.2]
Statistical Analysis 3: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 1.0000, Chan and Zhang Exact Method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-10.8 to 10.8]
Statistical Analysis 4: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0708, Chan and Zhang Exact Method; Risk Difference (RD) = 11.3, 90% CI 2-sided [-1.4 to 25.0]
Statistical Analysis 5: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0122, Chan and Zhang Exact Method; Risk Difference (RD) = 13.9, 90% CI 2-sided [4.7 to 27.0]
Statistical Analysis 6: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 1: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0016, Chan and Zhang Exact Method; Risk Difference (RD) = 21.6, 90% CI 2-sided [11.0 to 35.6]
Statistical Analysis 7: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.3950, Chan and Zhang Exact Method; Risk Difference (RD) = 2.7, 90% CI 2-sided [-9.8 to 16.1]
Statistical Analysis 8: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0173, Chan and Zhang Exact Method; Risk Difference (RD) = 19.7, 90% CI 2-sided [4.2 to 35.6]
Statistical Analysis 9: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0327, Chan and Zhang Exact Method; Risk Difference (RD) = 16.2, 90% CI 2-sided [1.4 to 31.0]
Statistical Analysis 10: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0011, Chan and Zhang Exact Method; Risk Difference (RD) = 30.8, 90% CI 2-sided [13.2 to 46.6]
Statistical Analysis 11: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1348, Chan and Zhang Exact Method; Risk Difference (RD) = 11.1, 90% CI 2-sided [-5.0 to 27.2]
Statistical Analysis 12: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 2: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0328, Chan and Zhang Exact Method; Risk Difference (RD) = 18.5, 90% CI 2-sided [1.5 to 34.8]
Statistical Analysis 13: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0769, Chan and Zhang Exact Method; Risk Difference (RD) = 10.8, 90% CI 2-sided [-1.8 to 24.4]
Statistical Analysis 14: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0005, Chan and Zhang Exact Method; Risk Difference (RD) = 30.7, 90% CI 2-sided [13.2 to 46.0]
Statistical Analysis 15: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p < 0.0001, Chan and Zhang Exact Method; Risk Difference (RD) = 37.8, 90% CI 2-sided [22.1 to 53.1]
Statistical Analysis 16: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0001, Chan and Zhang Exact Method; Risk Difference (RD) = 36.3, 90% CI 2-sided [19.7 to 51.8]
Statistical Analysis 17: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 1.0000, Chan and Zhang Exact Method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-16.5 to 16.5]
Statistical Analysis 18: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 3: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0173, Chan and Zhang Exact Method; Risk Difference (RD) = 23.8, 90% CI 2-sided [4.5 to 41.5]
Statistical Analysis 19: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.5663, Chan and Zhang Exact Method; Risk Difference (RD) = -2.7, 90% CI 2-sided [-19.9 to 14.2]
Statistical Analysis 20: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1243, Chan and Zhang Exact Method; Risk Difference (RD) = 14.6, 90% CI 2-sided [-3.8 to 32.6]
Statistical Analysis 21: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0460, Chan and Zhang Exact Method; Risk Difference (RD) = 18.9, 90% CI 2-sided [-0.5 to 36.6]
Statistical Analysis 22: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0130, Chan and Zhang Exact Method; Risk Difference (RD) = 25.7, 90% CI 2-sided [4.8 to 43.3]
Statistical Analysis 23: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1194, Chan and Zhang Exact Method; Risk Difference (RD) = 13.9, 90% CI 2-sided [-4.2 to 31.4]
Statistical Analysis 24: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 4: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0097, Chan and Zhang Exact Method; Risk Difference (RD) = 26.4, 90% CI 2-sided [6.5 to 44.4]
Statistical Analysis 25: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.1% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.5556, Chan and Zhang Exact Method; Risk Difference (RD) = -2.7, 90% CI 2-sided [-21.0 to 16.1]
Statistical Analysis 26: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 0.3% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0761, Chan and Zhang Exact Method; Risk Difference (RD) = 17.6, 90% CI 2-sided [-2.5 to 36.5]
Statistical Analysis 27: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 1.0% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0583, Chan and Zhang Exact Method; Risk Difference (RD) = 18.9, 90% CI 2-sided [-0.8 to 37.6]
Statistical Analysis 28: Comparison: Vehicle Cream Once Daily (QD) vs PF-06700841 3.0% Cream QD; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.1245, Chan and Zhang Exact Method; Risk Difference (RD) = 14.9, 90% CI 2-sided [-5.0 to 33.7]
Statistical Analysis 29: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 0.3% Cream BID; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0382, Chan and Zhang Exact Method; Risk Difference (RD) = 19.4, 90% CI 2-sided [1.5 to 36.5]
Statistical Analysis 30: Comparison: Vehicle Cream Twice Daily (BID) vs PF-06700841 1.0% Cream BID; At Week 6: Risk difference = difference in percentage of participants; Test type: Superiority; p = 0.0011, Chan and Zhang Exact Method; Risk Difference (RD) = 34.7, 90% CI 2-sided [13.2 to 51.4]

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent were events between first dose of investigational product and up to 28 days after the last dose of investigational product that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and all non-SAEs.
Time Frame: Baseline (Day 1) up to at least 28 days after last dose of study drug (approximately up to Week 11)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Participants
  TEAEs | 18 | 17 | 11 | 12 | 10 | 17 | 9 | 14
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Pre-defined Criteria For Vital Signs
Description: Pre-defined criteria included: 1) Diastolic blood pressure (DBP), a) sitting DBP: change of >= 20 millimeter of mercury (mmHg) increase, b) sitting DBP: change of >=20mmHg decrease, c) supine DBP: less than (<) 50 mmHg, d) supine DBP: change of >= 20mmHg increase, e) supine DBP: change of >= 20mmHg decrease; 2) Systolic blood pressure (SBP), a) sitting SBP: <90 mmHg, b) sitting SBP: change of >=30mmHg increase, c) sitting SBP: change of >=30mmHg decrease, d) supine SBP: change of >=30mmHg increase, e) supine SBP: change of >=30mmHg decrease and f) Supine SBP: value <90mmHg.
Time Frame: Baseline up to Week 6
Population: Safety analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the each specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 21 | 20 | 25 | 18 | 21 | 19 | 22 | 22
Participants
  Sitting DBP: Change >= 20 mm Hg increase: number analyzed (Participants) | 12 | 13 | 9 | 15 | 12 | 7 | 12 | 11
  Sitting DBP: Change >= 20 mm Hg increase | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Sitting DBP: Change >= 20mmHg decrease: number analyzed (Participants) | 12 | 13 | 9 | 15 | 12 | 7 | 12 | 11
  Sitting DBP: Change >= 20mmHg decrease | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Supine DBP: Value <50 mmHg | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Supine DBP: Change >= 20mmHg increase | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0
  Supine DBP: Change >= 20mmHg decrease | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Sitting SBP: <90mmHg: number analyzed (Participants) | 12 | 13 | 9 | 15 | 12 | 7 | 12 | 11
  Sitting SBP: <90mmHg | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Sitting SBP: change >= 30mmHg increase: number analyzed (Participants) | 12 | 13 | 9 | 15 | 12 | 7 | 12 | 11
  Sitting SBP: change >= 30mmHg increase | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Sitting SBP: change >= 30mmHg decrease: number analyzed (Participants) | 12 | 13 | 9 | 15 | 12 | 7 | 12 | 11
  Sitting SBP: change >= 30mmHg decrease | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Supine SBP: Change >= 30mmHg increase | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
  Supine SBP: Change >= 30mmHg decrease | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Supine SBP: Value <90mmHg | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Hemoglobin (HGB),hematocrit,erythrocytes (ery.),HDL cholesterol (chl.)<0.8*lower limit of normal(LLN);reticulocytes (ret.), ret./ery. (%)<0.5*LLN,>1.5*upper limit of normal (ULN);ery. mean corpuscular (EMC) volume,EMC HGB,EMC HGB concentration,potassium,chloride,calcium,bicarbonate<0.9*LLN,>1.1*ULN;platelets<0.5*LLN,>1.75*ULN;leukocytes (leu.),glucose<0.6*LLN,>1.5*ULN;lymphocytes (lym.), lym./leu.(%), neutrophils (neu.), neu./leu. (%), protein,albumin <0.8*LLN,>1.2*ULN;basophils (bas.), bas./leu.(%), eosinophils (eos.), eos./leu., monocytes (mon.), mon./leu.(%), urate >1.2*ULN;bilirubin (total, direct, indirect)>1.5*ULN;aspartate/alanine aminotransferase, gamma glutamyl transferase, lactate dehydrogenase, alkaline phosphatase>3.0*ULN;urea nitrogen, creatinine, triglycerides, chl.>1.3*ULN; sodium <0.95*LLN,>1.05*ULN; creatine kinase >2.0*ULN;Urine: pH<4.5,>8;glucose, ketones, protein, HGB, urobilinogen,bilirubin,nitrite,leukocyte esterase>=1;ery., leu.>= 20;hyaline casts>1;bacteria>20.
Time Frame: Baseline (Day 1) up to at least 28 days after last dose of study drug (approximately up to Week 11)
Population: Safety analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 35 | 35 | 37 | 35 | 36 | 36 | 36
Participants | 26 | 22 | 23 | 22 | 16 | 21 | 24 | 24

11. Secondary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings
Description: Clinically significant ECG criteria included PR interval: value greater than (>) 280 millisecond (msec), percentage change greater than equal to (>=) 25/50 percentage, QRS interval: value >120 msec, percentage change >= 50% and QT interval corrected using the Fridericia's formula (QTCF) value 450 msec and 30<=change<60.
Time Frame: Baseline up to Week 6
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 8 | 6 | 7 | 9 | 10 | 6 | 7 | 7
Participants
  PR interval : value >280 msec | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PR interval : %change>=25/50% | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
  QRS interval: value >120 msec | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  QRS interval: %Change>=50% | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  QTCF: 450 msec | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  QTCF: 30<=Change<60 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0

12. Secondary Outcome: Change From Baseline in Clinical Chemistry-Lactate Dehydrogenase Laboratory Values at Weeks 1, 2, 4, 6 and Follow-up Visit
Time Frame: Baseline, Weeks 1, 2, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 32 | 32 | 32 | 33 | 32 | 32 | 34 | 33
Units per liter
  Change at week 1: number analyzed (Participants) | 32 | 32 | 32 | 30 | 32 | 32 | 34 | 33
  Change at week 1 | 0.4 (25.99) | -7.4 (30.20) | -5.3 (16.99) | -9.3 (22.65) | -18.4 (33.42) | -8.0 (34.51) | -8.0 (19.37) | -4.3 (29.08)
  Change at week 2: number analyzed (Participants) | 32 | 27 | 30 | 33 | 27 | 28 | 31 | 30
  Change at week 2 | -8.8 (21.56) | -7.8 (27.99) | -1.9 (18.18) | -8.8 (23.70) | -15.8 (42.19) | -0.3 (22.81) | -8.0 (22.31) | -4.9 (24.49)
  Change at week 4: number analyzed (Participants) | 26 | 27 | 30 | 31 | 30 | 24 | 27 | 29
  Change at week 4 | -8.6 (23.93) | -5.4 (22.87) | -9.3 (19.61) | -12.1 (28.54) | -16.3 (33.97) | -1.0 (29.29) | -19.5 (19.94) | -3.7 (24.96)
  Change at week 6: number analyzed (Participants) | 30 | 26 | 31 | 31 | 28 | 23 | 31 | 32
  Change at week 6 | -8.8 (18.25) | -8.1 (32.02) | -1.5 (32.42) | -6.4 (28.53) | -18.2 (33.86) | -9.7 (20.68) | -11.2 (22.34) | -7.0 (24.65)
  Change at follow-up visit: number analyzed (Participants) | 26 | 28 | 31 | 30 | 27 | 30 | 30 | 26
  Change at follow-up visit | -12.3 (24.82) | -12.0 (28.83) | 4.0 (43.45) | -2.7 (26.27) | -15.1 (38.23) | -11.3 (29.39) | -13.3 (25.37) | 0.2 (16.48)

13. Secondary Outcome: Change From Baseline in Clinical Chemistry- Protein and Albumin Laboratory Values at Weeks 1, 2, 4, 6 and Follow-up Visit
Time Frame: Baseline, Weeks 1, 2, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Gram per deciliter
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 34 | 35 | 33 | 35 | 34 | 36 | 36 | 35
Gram per deciliter
  Protein: change at week 1: number analyzed (Participants) | 34 | 35 | 33 | 35 | 34 | 34 | 36 | 35
  Protein: change at week 1 | -0.01 (0.439) | -0.04 (0.294) | -0.14 (0.433) | -0.04 (0.264) | -0.03 (0.421) | -0.10 (0.360) | -0.01 (0.344) | -0.02 (0.301)
  Protein:change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Protein:change at week 2 | -0.09 (0.383) | 0.03 (0.303) | -0.18 (0.402) | -0.01 (0.275) | 0.01 (0.561) | 0.02 (0.503) | -0.04 (0.286) | -0.10 (0.299)
  Protein: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Protein: change at week 4 | -0.10 (0.380) | 0.07 (0.315) | -0.08 (0.429) | -0.03 (0.341) | -0.04 (0.465) | -0.18 (0.292) | -0.15 (0.242) | 0.03 (0.280)
  Protein: change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Protein: change at week 6 | -0.13 (0.403) | 0.13 (0.379) | -0.19 (0.452) | 0.01 (0.368) | -0.03 (0.405) | -0.10 (0.424) | -0.09 (0.368) | -0.09 (0.310)
  Protein: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Protein: change at follow-up visit | -0.07 (0.341) | 0.05 (0.457) | -0.15 (0.481) | -0.04 (0.404) | 0.03 (0.481) | -0.18 (0.471) | -0.09 (0.398) | 0.02 (0.299)
  Albumin:change at week 1: number analyzed (Participants) | 34 | 35 | 33 | 35 | 34 | 34 | 36 | 35
  Albumin:change at week 1 | -0.04 (0.269) | -0.05 (0.205) | -0.10 (0.283) | -0.02 (0.177) | 0.00 (0.256) | -0.05 (0.218) | -0.03 (0.246) | 0.00 (0.169)
  Albumin:change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Albumin:change at week 2 | -0.06 (0.235) | 0.02 (0.201) | -0.10 (0.256) | -0.02 (0.204) | -0.01 (0.283) | 0.02 (0.266) | -0.03 (0.174) | -0.06 (0.202)
  Albumin: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Albumin: change at week 4 | -0.08 (0.245) | 0.07 (0.172) | -0.08 (0.285) | 0.01 (0.239) | 0.04 (0.292) | -0.10 (0.232) | -0.08 (0.180) | 0.03 (0.224)
  Albumin:change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Albumin:change at week 6 | -0.08 (0.259) | 0.08 (0.245) | -0.14 (0.333) | -0.02 (0.269) | -0.00 (0.218) | -0.03 (0.252) | -0.07 (0.244) | -0.05 (0.227)
  Albumin: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Albumin: change at follow-up visit | -0.06 (0.247) | 0.10 (0.260) | -0.09 (0.277) | -0.04 (0.295) | -0.01 (0.346) | -0.09 (0.262) | -0.02 (0.211) | 0.06 (0.181)

14. Secondary Outcome: Change From Baseline in Clinical Chemistry- Urea Nitrogen, Urate, Calcium and Glucose Laboratory Values at Weeks 1, 2, 4, 6 and Follow-up Visit
Time Frame: Baseline, Weeks 1, 2, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Microgram per deciliter
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 34 | 35 | 33 | 35 | 34 | 34 | 36 | 35
Microgram per deciliter
  Urea nitrogen: change at week 1 | 0.9 (4.57) | 0.6 (3.04) | 0.1 (3.12) | 1.0 (3.19) | 1.0 (3.05) | 0.2 (2.19) | 0.4 (3.38) | -0.1 (2.65)
  Urea nitrogen: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Urea nitrogen: change at week 2 | 0.8 (3.89) | 0.0 (2.71) | 0.6 (3.54) | 0.9 (3.18) | 0.5 (3.63) | 0.6 (4.19) | 0.8 (2.99) | 0.4 (3.28)
  Urea nitrogen: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Urea nitrogen: change at week 4 | 0.6 (3.39) | 0.0 (3.04) | -0.0 (2.67) | 1.4 (3.06) | 0.5 (3.84) | -0.7 (2.96) | 1.3 (2.81) | -0.2 (3.61)
  Urea nitrogen: change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Urea nitrogen: change at week 6 | 0.7 (2.84) | -0.2 (3.11) | -0.6 (3.61) | 0.9 (3.27) | 0.3 (3.82) | -0.8 (3.24) | 0.2 (3.52) | -0.4 (3.69)
  Urea nitrogen: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Urea nitrogen: change at follow-up visit | 0.0 (3.17) | -0.3 (3.13) | 0.4 (2.60) | 1.2 (4.22) | 0.2 (2.87) | 0.8 (3.78) | 0.5 (3.42) | 0.1 (3.78)
  Urate:change at week 1 | 0.16 (0.807) | 0.01 (0.606) | 0.16 (0.678) | -0.01 (0.561) | 0.00 (0.739) | 0.05 (0.661) | -0.02 (0.704) | -0.14 (0.890)
  Urate: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Urate: change at week 2 | 0.30 (0.990) | -0.11 (0.655) | 0.12 (0.617) | -0.03 (0.649) | -0.15 (0.842) | 0.27 (1.025) | -0.03 (0.718) | -0.37 (1.059)
  Urate: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Urate: change at week 4 | 0.21 (0.497) | 0.14 (0.731) | 0.06 (0.756) | -0.06 (0.621) | -0.14 (0.856) | 0.22 (0.806) | -0.21 (0.663) | -0.16 (0.713)
  Urate: change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Urate: change at week 6 | 0.13 (0.728) | 0.07 (0.984) | -0.02 (0.831) | 0.06 (0.630) | -0.02 (0.649) | 0.06 (0.534) | -0.11 (0.827) | -0.21 (1.084)
  Urate: change at follow- up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Urate: change at follow- up visit | -0.11 (0.721) | -0.33 (0.753) | 0.05 (0.763) | -0.21 (0.554) | -0.02 (0.810) | 0.02 (0.590) | -0.08 (0.677) | -0.20 (0.989)
  Calcium:change at week 1 | 0.01 (0.419) | 0.01 (0.259) | -0.06 (0.377) | -0.02 (0.248) | 0.07 (0.386) | -0.02 (0.303) | -0.01 (0.295) | 0.09 (0.318)
  Calcium: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Calcium: change at week 2 | -0.08 (0.417) | 0.00 (0.268) | -0.10 (0.362) | 0.05 (0.296) | 0.07 (0.423) | 0.03 (0.389) | -0.10 (0.293) | -0.01 (0.244)
  Calcium: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Calcium: change at week 4 | -0.04 (0.354) | 0.11 (0.329) | -0.07 (0.345) | 0.05 (0.272) | 0.00 (0.376) | -0.08 (0.309) | -0.03 (0.257) | 0.10 (0.341)
  Calcium: change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Calcium: change at week 6 | -0.04 (0.355) | 0.10 (0.303) | -0.21 (0.393) | 0.03 (0.315) | 0.00 (0.397) | -0.05 (0.335) | -0.05 (0.464) | -0.04 (0.337)
  Calcium: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Calcium: change at follow-up visit | 0.00 (0.317) | -0.01 (0.345) | -0.08 (0.409) | 0.00 (0.323) | 0.10 (0.441) | -0.05 (0.419) | 0.01 (0.378) | 0.05 (0.356)
  Glucose:change at week 1: number analyzed (Participants) | 34 | 35 | 33 | 34 | 34 | 33 | 36 | 35
  Glucose:change at week 1 | 4.9 (8.73) | 5.7 (13.97) | 3.4 (14.62) | 4.5 (8.60) | 4.4 (16.14) | 4.5 (29.90) | 5.6 (13.14) | 3.3 (13.58)
  Glucose: change at week 2: number analyzed (Participants) | 33 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Glucose: change at week 2 | 9.7 (23.71) | 1.2 (17.34) | 0.6 (10.97) | 3.2 (12.63) | 3.1 (10.00) | -1.9 (13.51) | 7.9 (16.67) | 2.7 (18.07)
  Glucose: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Glucose: change at week 4 | 7.3 (15.60) | 0.5 (12.50) | -1.2 (15.86) | 4.5 (13.99) | 2.8 (20.20) | 1.3 (24.01) | 10.7 (26.13) | 3.4 (18.33)
  Glucose: change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Glucose: change at week 6 | 3.5 (9.19) | 2.4 (17.55) | -1.7 (10.62) | 2.1 (13.80) | -0.5 (9.77) | -3.4 (16.37) | 4.3 (12.23) | 1.5 (12.62)
  Glucose: change at follow -up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Glucose: change at follow -up visit | 4.5 (11.58) | 2.2 (11.45) | 4.8 (13.28) | 4.6 (14.77) | 6.0 (13.79) | 6.2 (16.75) | 9.1 (17.21) | 2.0 (22.43)

15. Secondary Outcome: Change From Baseline in Clinical Chemistry- Sodium, Potassium, Chloride and Bicarbonate Laboratory Values at Weeks 1, 2, 4, 6 and Follow-up Visit
Time Frame: Baseline, Weeks 1, 2, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Milliequivalents per liter
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 34 | 35 | 33 | 35 | 34 | 34 | 36 | 35
Milliequivalents per liter
  Sodium: change at week 1 | 0.1 (2.34) | -0.0 (1.77) | -0.7 (2.04) | -0.6 (2.17) | -0.4 (3.50) | 0.4 (1.97) | 0.0 (2.08) | -0.1 (3.39)
  Sodium: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Sodium: change at week 2 | -0.5 (2.23) | -0.3 (1.89) | -0.1 (2.39) | -0.2 (2.18) | -0.4 (3.61) | -0.2 (2.61) | -0.5 (2.20) | -0.3 (3.45)
  Sodium:change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Sodium:change at week 4 | -0.3 (2.70) | 0.6 (1.83) | -0.2 (2.44) | -0.7 (2.71) | -0.4 (3.08) | -0.4 (2.72) | -0.1 (1.77) | -0.3 (3.28)
  Sodium:change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Sodium:change at week 6 | -0.8 (2.31) | 0.0 (2.39) | -0.2 (2.23) | -0.9 (2.40) | -0.9 (3.55) | 0.9 (2.50) | -0.1 (2.23) | -0.5 (2.49)
  Sodium: change at follow up: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Sodium: change at follow up | -0.4 (3.26) | 0.5 (2.50) | -0.1 (2.45) | -0.3 (2.41) | -0.8 (3.59) | 0.7 (1.94) | -0.1 (2.46) | 0.1 (3.32)
  Potassium: change at week 1: number analyzed (Participants) | 34 | 35 | 33 | 35 | 34 | 34 | 36 | 34
  Potassium: change at week 1 | -0.00 (0.363) | 0.08 (0.282) | 0.03 (0.372) | 0.02 (0.347) | 0.07 (0.343) | 0.01 (0.337) | 0.00 (0.429) | 0.20 (0.464)
  Potassium:change at week 2: number analyzed (Participants) | 33 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Potassium:change at week 2 | -0.14 (0.367) | 0.04 (0.298) | -0.07 (0.338) | 0.04 (0.359) | 0.07 (0.346) | 0.00 (0.245) | -0.16 (0.438) | -0.02 (0.322)
  Potassium: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Potassium: change at week 4 | 0.01 (0.389) | -0.06 (0.285) | -0.02 (0.350) | -0.01 (0.327) | 0.05 (0.375) | -0.09 (0.300) | -0.03 (0.415) | 0.26 (0.350)
  Potassium: change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Potassium: change at week 6 | -0.09 (0.373) | 0.03 (0.295) | -0.06 (0.332) | 0.03 (0.407) | -0.06 (0.262) | -0.06 (0.309) | -0.10 (0.355) | 0.09 (0.388)
  Potassium: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Potassium: change at follow-up visit | -0.11 (0.379) | 0.10 (0.375) | 0.03 (0.394) | 0.04 (0.351) | 0.12 (0.358) | 0.05 (0.293) | -0.09 (0.475) | 0.26 (0.460)
  Chloride: change at week 1 | 0.1 (2.11) | 0.3 (1.86) | 0.3 (1.57) | 0.0 (2.54) | 0.0 (2.66) | 0.6 (2.11) | 0.5 (2.02) | 0.5 (2.83)
  Chloride: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 32
  Chloride: change at week 2 | -0.2 (2.52) | -0.2 (2.08) | 0.7 (2.03) | 0.2 (2.50) | -0.2 (2.87) | 0.4 (2.70) | 0.4 (2.15) | 0.2 (2.99)
  Chloride: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 31 | 30
  Chloride: change at week 4 | 0.3 (2.05) | 0.6 (1.89) | 0.2 (2.68) | -0.4 (2.23) | -0.3 (2.16) | 0.3 (3.28) | 1.0 (2.21) | -0.2 (2.57)
  Chloride:change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Chloride:change at week 6 | -0.6 (1.98) | 0.1 (2.27) | 0.0 (2.34) | -0.5 (2.44) | -0.4 (3.05) | 0.5 (2.93) | 0.9 (2.73) | 0.0 (2.32)
  Chloride: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Chloride: change at follow-up visit | 0.6 (2.97) | -0.3 (2.16) | 0.8 (2.64) | 0.1 (2.41) | -0.4 (2.90) | 1.3 (2.11) | 0.3 (2.35) | 0.4 (3.16)
  Bicarbonate: change at week 1: number analyzed (Participants) | 34 | 35 | 33 | 33 | 34 | 33 | 36 | 35
  Bicarbonate: change at week 1 | 0.13 (2.548) | -0.38 (1.759) | -0.20 (1.965) | -0.18 (1.768) | 0.28 (1.638) | 0.09 (2.209) | -0.21 (2.388) | -0.02 (1.651)
  Bicarbonate: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 31 | 30 | 33 | 32
  Bicarbonate: change at week 2 | 0.08 (2.229) | -0.40 (2.151) | -0.51 (1.956) | 0.10 (2.129) | -0.13 (1.931) | -0.15 (2.341) | -0.60 (2.354) | -0.07 (1.828)
  Bicarbonate: change at week 4: number analyzed (Participants) | 29 | 28 | 33 | 31 | 32 | 24 | 30 | 30
  Bicarbonate: change at week 4 | 0.21 (2.739) | 0.05 (2.128) | -0.24 (2.484) | 0.34 (1.868) | 0.02 (2.011) | 0.14 (1.286) | -0.00 (2.695) | 0.02 (1.704)
  Bicarbonate: change at week 6: number analyzed (Participants) | 30 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Bicarbonate: change at week 6 | 0.52 (2.560) | -0.44 (2.598) | 0.66 (2.132) | 0.27 (2.204) | 0.12 (2.407) | 0.63 (2.096) | -0.19 (2.038) | -0.20 (2.217)
  Bicarbonate: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 32 | 32 | 29 | 31 | 32 | 30
  Bicarbonate: change at follow-up visit | -0.02 (2.916) | 0.66 (2.209) | 0.41 (2.056) | 0.75 (2.386) | 0.43 (2.162) | 0.08 (1.643) | 0.18 (2.300) | 1.09 (2.049)

16. Secondary Outcome: Change From Baseline in Hematology- Hemoglobin Laboratory Values at Weeks 1, 2, 4, 6 and Follow-up Visit
Time Frame: Baseline, Weeks 1, 2, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Gram per deciliter
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 34 | 37 | 33 | 34 | 34 | 33 | 35 | 34
Gram per deciliter
  Change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Change at week 1 | -0.01 (0.790) | -0.22 (0.620) | -0.36 (0.775) | -0.12 (0.678) | -0.26 (0.726) | -0.19 (0.698) | -0.21 (0.584) | -0.27 (0.679)
  Change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Change at week 2 | -0.16 (0.636) | -0.09 (0.566) | -0.64 (0.715) | -0.24 (0.657) | -0.22 (0.798) | -0.16 (0.830) | -0.25 (0.625) | -0.32 (0.793)
  Change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Change at week 4 | 0.03 (0.725) | -0.17 (0.630) | -0.48 (0.659) | -0.25 (0.628) | -0.06 (0.821) | -0.27 (0.789) | -0.32 (0.701) | -0.20 (0.658)
  Change at week 6: number analyzed (Participants) | 29 | 37 | 31 | 32 | 31 | 24 | 32 | 33
  Change at week 6 | -0.13 (0.832) | -0.06 (0.614) | -0.48 (0.767) | -0.03 (0.617) | -0.11 (0.775) | -0.22 (0.724) | -0.21 (0.833) | -0.28 (0.683)
  Change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 30 | 30
  Change at follow-up visit | 0.05 (0.613) | -0.04 (0.717) | -0.49 (0.777) | -0.09 (0.784) | 0.00 (0.773) | -0.27 (0.756) | -0.12 (0.826) | -0.18 (0.740)

17. Secondary Outcome: Change From Baseline in Hematology - Hematocrit, Reticulocytes/Erythrocytes, Lymphocytes/Leukocytes, Neutrophils/Leukocytes, Basophils/Leukocytes, Eosinophils/Leukocytes and Monocytes/Leukocytes Laboratory Values at Weeks 1, 2, 4, 6 and Follow-up Visit
Time Frame: Baseline, Weeks 1, 2, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 34 | 35 | 33 | 34 | 34 | 33 | 35 | 34
Percentage of cells
  Hematocrit: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 33
  Hematocrit: change at week 1 | 0.2 (2.51) | -0.8 (2.11) | -1.3 (2.61) | -0.4 (2.27) | -0.8 (2.41) | -0.5 (1.97) | -0.9 (2.04) | -0.9 (2.30)
  Hematocrit: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 30
  Hematocrit: change at week 2 | -0.5 (2.19) | -0.8 (2.12) | -1.8 (2.42) | -0.9 (2.32) | -0.7 (2.58) | -0.9 (2.55) | -0.7 (2.24) | -1.0 (2.61)
  Hematocrit: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 30 | 31 | 25 | 30 | 30
  Hematocrit: change at week 4 | 0.0 (2.45) | -0.8 (1.96) | -1.8 (2.06) | -0.8 (2.34) | 0.0 (2.73) | -1.0 (2.34) | -0.9 (2.29) | -0.5 (2.56)
  Hematocrit: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Hematocrit: change at week 6 | -0.6 (2.47) | -0.9 (1.93) | -1.6 (2.64) | -0.7 (2.23) | -0.6 (2.51) | -1.1 (1.98) | -1.1 (2.84) | -0.8 (2.60)
  Hematocrit: change at follow-up (FU) visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Hematocrit: change at follow-up (FU) visit | 0.3 (2.49) | -0.7 (2.24) | -1.4 (3.05) | -0.7 (2.39) | -0.2 (2.50) | -0.6 (2.20) | -0.6 (2.73) | -0.3 (2.78)
  Reticulocytes/Erythrocytes change at week 1: number analyzed (Participants) | 31 | 31 | 29 | 29 | 27 | 28 | 31 | 27
  Reticulocytes/Erythrocytes change at week 1 | 0.03 (0.317) | 0.14 (0.378) | 0.02 (0.483) | 0.06 (0.364) | 0.11 (0.318) | 0.01 (0.320) | 0.04 (0.355) | 0.01 (0.329)
  Reticulocytes/Erythrocytes: change at week 2: number analyzed (Participants) | 31 | 30 | 29 | 29 | 25 | 26 | 29 | 24
  Reticulocytes/Erythrocytes: change at week 2 | -0.03 (0.382) | 0.17 (0.325) | 0.09 (0.413) | -0.02 (0.473) | 0.19 (0.443) | -0.10 (0.318) | 0.06 (0.315) | -0.01 (0.389)
  Reticulocytes/Erythrocytes: change at week 4: number analyzed (Participants) | 25 | 24 | 30 | 27 | 25 | 23 | 26 | 23
  Reticulocytes/Erythrocytes: change at week 4 | 0.16 (0.596) | -0.08 (0.359) | 0.01 (0.460) | 0.19 (0.429) | 0.10 (0.409) | 0.03 (0.290) | 0.04 (0.446) | 0.05 (0.374)
  Reticulocytes/Erythrocytes: change at week 6: number analyzed (Participants) | 26 | 25 | 28 | 28 | 24 | 22 | 28 | 26
  Reticulocytes/Erythrocytes: change at week 6 | -0.06 (0.382) | 0.02 (0.361) | 0.02 (0.473) | 0.01 (0.486) | 0.15 (0.399) | -0.15 (0.310) | -0.01 (0.355) | 0.01 (0.463)
  Reticulocytes/Erythrocytes:change at FU visit: number analyzed (Participants) | 27 | 25 | 27 | 27 | 23 | 27 | 27 | 23
  Reticulocytes/Erythrocytes:change at FU visit | -0.11 (0.396) | -0.02 (0.384) | 0.10 (0.435) | -0.10 (0.398) | -0.03 (0.298) | -0.09 (0.331) | -0.19 (0.395) | 0.11 (0.448)
  Lymphocytes/Leukocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Lymphocytes/Leukocytes: change at week 1 | -0.43 (6.772) | 0.68 (5.814) | 2.33 (5.616) | 0.06 (4.765) | 1.31 (6.259) | 0.59 (5.179) | 0.49 (5.509) | 1.79 (6.269)
  Lymphocytes/Leukocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Lymphocytes/Leukocytes: change at week 2 | 0.20 (6.175) | 0.84 (7.544) | 1.68 (5.208) | 1.50 (5.639) | 0.23 (6.175) | 0.50 (5.405) | 0.72 (6.638) | 0.86 (7.264)
  Lymphocytes/Leukocytes: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Lymphocytes/Leukocytes: change at week 4 | 1.58 (7.591) | 0.51 (7.297) | 1.43 (5.298) | 0.43 (7.586) | 2.41 (6.577) | -1.38 (5.415) | 1.07 (5.739) | 0.56 (7.264)
  Lymphocytes/Leukocytes: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Lymphocytes/Leukocytes: change at week 6 | -0.92 (6.701) | -0.06 (5.461) | 0.82 (6.685) | 1.28 (5.881) | 1.65 (5.818) | 0.50 (4.452) | -0.04 (5.300) | 1.52 (7.266)
  Lymphocytes/Leukocytes: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Lymphocytes/Leukocytes: change at follow-up visit | 1.53 (6.219) | 1.25 (4.974) | 1.61 (6.597) | -0.85 (6.367) | 1.34 (6.165) | 0.22 (6.315) | 0.07 (5.103) | 2.48 (6.914)
  Neutrophils/Leukocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Neutrophils/Leukocytes: change at week 1 | 0.57 (7.515) | -0.95 (6.957) | -2.93 (6.191) | 0.30 (5.755) | -0.96 (7.843) | -0.17 (5.769) | -1.87 (6.873) | -1.44 (6.580)
  Neutrophils/Leukocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Neutrophils/Leukocytes: change at week 2 | -0.12 (7.827) | -0.34 (8.219) | -1.70 (6.037) | -1.50 (6.578) | -0.24 (6.146) | -0.49 (6.665) | -1.04 (7.376) | -0.56 (8.017)
  Neutrophils/Leukocytes: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Neutrophils/Leukocytes: change at week 4 | -1.42 (8.812) | -0.30 (7.754) | -1.52 (6.661) | 0.06 (8.536) | -2.25 (7.468) | 1.65 (6.622) | -1.42 (6.498) | -0.45 (7.362)
  Neutrophils/Leukocytes: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Neutrophils/Leukocytes: change at week 6 | 0.95 (8.648) | -0.58 (7.009) | -0.64 (6.833) | -1.14 (6.872) | -1.15 (6.969) | -0.56 (5.699) | 0.13 (6.029) | -1.01 (8.445)
  Neutrophils/Leukocytes: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Neutrophils/Leukocytes: change at follow-up visit | -1.71 (7.046) | -0.65 (6.057) | -1.86 (6.892) | 1.32 (7.355) | -1.32 (6.559) | -0.41 (6.961) | -0.71 (6.590) | -2.04 (7.700)
  Basophils/Leukocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Basophils/Leukocytes: change at week 1 | -0.06 (0.431) | -0.02 (0.690) | -0.06 (0.524) | 0.08 (0.319) | 0.03 (0.515) | -0.03 (0.291) | -0.01 (0.411) | -0.01 (0.570)
  Basophils/Leukocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Basophils/Leukocytes: change at week 2 | -0.02 (0.304) | 0.01 (0.493) | -0.09 (0.342) | 0.02 (0.323) | -0.03 (0.532) | 0.03 (0.355) | -0.06 (0.624) | -0.24 (0.709)
  Basophils/Leukocytes: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Basophils/Leukocytes: change at week 4 | -0.07 (0.485) | 0.06 (0.651) | -0.03 (0.420) | 0.01 (0.402) | -0.08 (0.712) | -0.05 (0.362) | -0.01 (0.465) | -0.10 (0.464)
  Basophils/Leukocytes: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Basophils/Leukocytes: change at week 6 | -0.07 (0.272) | 0.11 (0.809) | -0.12 (0.480) | 0.08 (0.458) | -0.16 (0.557) | -0.05 (0.296) | -0.12 (0.576) | -0.17 (0.750)
  Basophils/Leukocytes: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Basophils/Leukocytes: change at follow-up visit | -0.04 (0.360) | -0.15 (0.476) | -0.13 (0.443) | 0.02 (0.512) | -0.25 (0.541) | -0.05 (0.449) | 0.01 (0.472) | -0.25 (0.572)
  Eosinophils/Leukocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Eosinophils/Leukocytes: change at week 1 | -0.09 (1.390) | 0.17 (1.840) | 0.17 (0.934) | -0.37 (1.549) | -0.31 (1.607) | -0.19 (1.410) | 0.89 (1.850) | -0.23 (1.339)
  Eosinophils/Leukocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Eosinophils/Leukocytes: change at week 2 | -0.11 (1.801) | -0.20 (1.298) | -0.16 (1.284) | 0.11 (1.460) | -0.27 (1.131) | -0.14 (1.199) | 0.16 (1.304) | -0.05 (1.531)
  Eosinophils/Leukocytes: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Eosinophils/Leukocytes: change at week 4 | 0.42 (1.982) | -0.12 (1.725) | 0.15 (1.884) | -0.37 (1.729) | -0.35 (1.431) | -0.34 (1.258) | 0.40 (1.468) | -0.37 (1.747)
  Eosinophils/Leukocytes: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Eosinophils/Leukocytes: change at week 6 | -0.03 (1.522) | 0.22 (1.570) | -0.04 (1.213) | 0.02 (2.126) | -0.15 (1.714) | -0.01 (1.767) | 0.05 (1.229) | -0.19 (1.840)
  Eosinophils/Leukocytes: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Eosinophils/Leukocytes: change at follow-up visit | 0.16 (1.754) | -0.24 (1.860) | -0.09 (1.155) | -0.41 (2.188) | 0.12 (1.954) | -0.05 (2.805) | 0.50 (1.986) | -0.13 (2.021)
  Monocytes/Leukocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Monocytes/Leukocytes: change at week 1 | 0.02 (1.913) | 0.12 (1.391) | 0.50 (1.428) | -0.06 (1.409) | -0.01 (1.593) | -0.19 (1.043) | 0.51 (1.275) | -0.11 (1.251)
  Monocytes/Leukocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Monocytes/Leukocytes: change at week 2 | 0.04 (2.055) | -0.31 (1.502) | 0.30 (1.522) | -0.13 (1.267) | 0.38 (1.362) | 0.11 (1.318) | 0.22 (1.414) | -0.01 (1.755)
  Monocytes/Leukocytes : change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Monocytes/Leukocytes : change at week 4 | -0.51 (2.509) | -0.17 (1.966) | -0.02 (2.072) | -0.10 (1.582) | 0.22 (1.323) | 0.14 (1.323) | -0.03 (1.039) | 0.33 (1.695)
  Monocytes/Leukocytes : change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Monocytes/Leukocytes : change at week 6 | 0.06 (2.488) | 0.33 (2.257) | -0.00 (1.813) | -0.24 (1.217) | -0.12 (1.030) | 0.13 (0.807) | -0.02 (1.324) | -0.16 (1.516)
  Monocytes/Leukocytes : change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Monocytes/Leukocytes : change at follow-up visit | 0.06 (2.105) | -0.22 (1.304) | 0.50 (1.463) | -0.07 (1.226) | 0.13 (1.205) | 0.26 (1.543) | 0.15 (1.599) | -0.04 (1.047)

18. Secondary Outcome: Change From Baseline in Hematology- Erythrocytes and Reticulocytes Laboratory Values at Weeks 1, 2, 4, 6 and Follow-up Visit
Time Frame: Baseline, Weeks 1, 2, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 10^12*cells per liter
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 34 | 35 | 33 | 34 | 34 | 33 | 35 | 34
10^12*cells per liter
  Erythrocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Erythrocytes: change at week 1 | 0.03 (0.261) | -0.07 (0.232) | -0.12 (0.264) | -0.04 (0.252) | -0.08 (0.254) | -0.08 (0.298) | -0.08 (0.192) | -0.09 (0.240)
  Erythrocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Erythrocytes: change at week 2 | -0.05 (0.234) | -0.03 (0.212) | -0.18 (0.251) | -0.10 (0.208) | -0.07 (0.242) | -0.10 (0.366) | -0.06 (0.229) | -0.11 (0.232)
  Erythrocytes: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Erythrocytes: change at week 4 | -0.01 (0.216) | -0.05 (0.221) | -0.16 (0.251) | -0.10 (0.233) | 0.01 (0.275) | -0.12 (0.271) | -0.08 (0.248) | -0.06 (0.219)
  Erythrocytes: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Erythrocytes: change at week 6 | -0.04 (0.247) | -0.01 (0.180) | -0.17 (0.265) | -0.04 (0.238) | -0.02 (0.262) | -0.10 (0.256) | -0.07 (0.303) | -0.08 (0.239)
  Erythrocytes: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Erythrocytes: change at follow-up visit | 0.03 (0.220) | 0.02 (0.244) | -0.15 (0.266) | -0.03 (0.254) | 0.04 (0.300) | -0.08 (0.280) | -0.03 (0.308) | -0.05 (0.262)
  Reticulocytes: change at week 1: number analyzed (Participants) | 31 | 31 | 29 | 29 | 27 | 28 | 31 | 27
  Reticulocytes: change at week 1 | 0.0 (0.02) | 0.0 (0.02) | -0.0 (0.02) | 0.0 (0.02) | 0.0 (0.02) | 0.0 (0.01) | 0.0 (0.02) | -0.0 (0.02)
  Reticulocytes: change at week 2: number analyzed (Participants) | 31 | 30 | 29 | 29 | 25 | 26 | 29 | 24
  Reticulocytes: change at week 2 | -0.0 (0.02) | 0.0 (0.02) | 0.0 (0.02) | -0.0 (0.02) | 0.0 (0.02) | -0.0 (0.02) | 0.0 (0.02) | -0.0 (0.02)
  Reticulocytes: change at week 4: number analyzed (Participants) | 25 | 24 | 30 | 27 | 25 | 23 | 26 | 23
  Reticulocytes: change at week 4 | 0.0 (0.03) | -0.0 (0.02) | -0.0 (0.02) | 0.0 (0.02) | 0.0 (0.02) | -0.0 (0.01) | -0.0 (0.02) | 0.0 (0.02)
  Reticulocytes: change at week 6: number analyzed (Participants) | 26 | 25 | 28 | 28 | 24 | 22 | 28 | 26
  Reticulocytes: change at week 6 | -0.0 (0.02) | 0.0 (0.02) | 0.0 (0.02) | -0.0 (0.02) | 0.0 (0.02) | -0.0 (0.01) | -0.0 (0.02) | 0.0 (0.02)
  Reticulocytes: change at follow-up visit: number analyzed (Participants) | 27 | 25 | 27 | 27 | 23 | 27 | 27 | 23
  Reticulocytes: change at follow-up visit | -0.0 (0.02) | -0.0 (0.02) | 0.0 (0.02) | -0.0 (0.02) | -0.0 (0.01) | -0.0 (0.02) | -0.0 (0.02) | 0.0 (0.02)

19. Secondary Outcome: Change From Baseline in Hematology- Platelets, Leukocytes, Lymphocytes, Neutrophils, Basophils, Eosinophils and Monocytes Laboratory Values at Weeks 1, 2, 4, 6 and Follow-up Visit
Time Frame: Baseline, Weeks 1, 2, 4, 6 and follow up visit (28 days after last dose of study drug = maximum up to Day 71)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 10^9 *cells per liter
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 34 | 35 | 33 | 34 | 34 | 33 | 35 | 34
10^9 *cells per liter
  Platelets: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Platelets: change at week 1 | 0.9 (60.03) | 6.8 (34.08) | -3.3 (32.39) | 1.0 (25.76) | 8.5 (41.61) | 6.6 (33.40) | -2.1 (31.94) | 12.6 (44.08)
  Platelets: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Platelets: change at week 2 | -4.9 (58.16) | 7.1 (43.34) | -8.1 (41.92) | -0.1 (32.45) | 5.0 (31.39) | -4.9 (31.84) | 7.5 (37.94) | 14.8 (50.99)
  Platelets: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Platelets: change at week 4 | 10.5 (36.42) | 10.1 (37.55) | -2.4 (37.68) | -0.3 (36.27) | -5.9 (37.47) | 4.4 (37.79) | 0.7 (36.51) | 11.0 (46.26)
  Platelets: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Platelets: change at week 6 | 4.9 (35.17) | -3.3 (32.76) | -6.6 (41.66) | -2.3 (32.70) | -5.2 (38.53) | 0.2 (37.28) | -1.8 (37.05) | 8.6 (47.85)
  Platelets: change at follow-up visit: number analyzed (Participants) | 29 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Platelets: change at follow-up visit | 1.3 (30.48) | 16.3 (37.13) | -8.5 (30.15) | 0.1 (32.36) | 10.2 (47.30) | -5.2 (40.70) | 5.8 (48.55) | 2.5 (58.75)
  Leukocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Leukocytes: change at week 1 | 0.027 (1.8740) | 0.395 (1.0940) | -0.051 (1.2403) | 0.407 (1.2225) | 0.259 (1.1290) | 0.068 (1.2929) | 0.238 (1.4993) | -0.025 (2.3529)
  Leukocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 31 | 33
  Leukocytes: change at week 2 | -0.206 (1.8886) | 0.459 (1.5567) | -0.288 (1.6842) | -0.094 (1.2877) | -0.116 (1.0364) | -0.007 (1.2637) | 0.422 (1.8986) | -0.006 (2.3428)
  Leukocytes: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Leukocytes: change at week 4 | -0.203 (1.7390) | 0.729 (1.3199) | 0.189 (1.3534) | 0.085 (1.3541) | -0.074 (1.0641) | 0.398 (1.5999) | 0.168 (1.0902) | 0.041 (2.1647)
  Leukocytes: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Leukocytes: change at week 6 | 0.160 (1.7059) | 0.066 (1.0672) | -0.505 (1.6474) | 0.237 (1.4501) | -0.244 (1.2763) | -0.269 (1.0761) | -0.048 (1.3823) | -0.347 (2.1442)
  Leukocytes: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Leukocytes: change at follow-up visit | -0.066 (1.5744) | 0.479 (1.0939) | -0.048 (2.0206) | 0.329 (1.3938) | 0.123 (0.8496) | -0.117 (1.4856) | 0.210 (1.7456) | -0.404 (2.4817)
  Lymphocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Lymphocytes: change at week 1 | -0.008 (0.5539) | 0.124 (0.3659) | 0.107 (0.3130) | 0.081 (0.3839) | 0.186 (0.3840) | 0.051 (0.3557) | 0.089 (0.4320) | 0.223 (0.3849)
  Lymphocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Lymphocytes: change at week 2 | -0.061 (0.5558) | 0.145 (0.3735) | 0.010 (0.4115) | 0.044 (0.4225) | 0.012 (0.4251) | -0.003 (0.3165) | 0.070 (0.4603) | 0.169 (0.5319)
  Lymphocytes: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Lymphocytes: change at week 4 | 0.107 (0.4302) | 0.229 (0.3998) | 0.135 (0.4400) | 0.012 (0.4596) | 0.139 (0.3977) | 0.039 (0.4169) | 0.127 (0.2630) | 0.176 (0.6274)
  Lymphocytes: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Lymphocytes: change at week 6 | 0.033 (0.3375) | 0.016 (0.3437) | -0.079 (0.4826) | 0.104 (0.4337) | 0.068 (0.3168) | -0.033 (0.3092) | 0.027 (0.2455) | 0.079 (0.3846)
  Lymphocytes: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Lymphocytes: change at follow-up visit | 0.134 (0.3256) | 0.194 (0.3533) | 0.065 (0.6042) | -0.022 (0.4419) | 0.130 (0.4277) | -0.035 (0.4054) | 0.050 (0.4699) | 0.195 (0.4663)
  Neutrophils: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Neutrophils: change at week 1 | 0.027 (1.6137) | 0.205 (0.9185) | -0.177 (1.0805) | 0.319 (1.0276) | 0.069 (1.0706) | 0.017 (1.1291) | 0.030 (1.3015) | -0.251 (2.2421)
  Neutrophils: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Neutrophils: change at week 2 | -0.119 (1.5672) | 0.293 (1.5459) | -0.261 (1.3969) | -0.136 (1.0669) | -0.109 (0.9653) | -0.015 (1.1305) | 0.288 (1.7822) | -0.190 (2.0749)
  Neutrophils: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Neutrophils: change at week 4 | -0.304 (1.6117) | 0.441 (1.2814) | 0.036 (1.1595) | 0.096 (1.3199) | -0.190 (1.0404) | 0.338 (1.3577) | -0.005 (0.9958) | -0.158 (2.0005)
  Neutrophils: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Neutrophils: change at week 6 | 0.112 (1.6282) | -0.001 (0.8996) | -0.362 (1.3154) | 0.112 (1.2240) | -0.250 (1.1720) | -0.228 (0.9681) | -0.064 (1.2422) | -0.376 (2.1125)
  Neutrophils: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Neutrophils: change at follow-up visit | -0.229 (1.3379) | 0.261 (0.8874) | -0.114 (1.4545) | 0.343 (1.3049) | -0.020 (0.7731) | -0.093 (1.2340) | 0.088 (1.4614) | -0.562 (2.3227)
  Basophils: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Basophils: change at week 1 | -0.006 (0.0319) | 0.004 (0.0445) | -0.007 (0.0349) | 0.010 (0.0258) | 0.003 (0.0361) | 0.001 (0.0191) | 0.002 (0.0299) | 0.002 (0.0343)
  Basophils: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Basophils: change at week 2 | -0.002 (0.0179) | 0.004 (0.0261) | -0.009 (0.0276) | 0.001 (0.0197) | -0.005 (0.0394) | 0.003 (0.0244) | -0.003 (0.0433) | -0.012 (0.0428)
  Basophils: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Basophils: change at week 4 | -0.006 (0.0328) | 0.011 (0.0404) | -0.002 (0.0300) | 0.001 (0.0256) | -0.007 (0.0495) | -0.001 (0.0255) | -0.001 (0.0337) | -0.004 (0.0323)
  Basophils: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Basophils: change at week 6 | -0.005 (0.0186) | 0.009 (0.0489) | -0.012 (0.0313) | 0.008 (0.0344) | -0.015 (0.0415) | -0.004 (0.0188) | -0.009 (0.0373) | -0.015 (0.0383)
  Basophils: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Basophils: change at follow-up visit | -0.004 (0.0265) | -0.003 (0.0259) | -0.007 (0.0321) | 0.007 (0.0407) | -0.015 (0.0426) | -0.005 (0.0269) | 0.001 (0.0295) | -0.019 (0.0361)
  Eosinophils: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Eosinophils: change at week 1 | 0.007 (0.0964) | 0.036 (0.0963) | -0.004 (0.1092) | -0.011 (0.0930) | -0.014 (0.1216) | -0.008 (0.1148) | 0.068 (0.0959) | -0.006 (0.1165)
  Eosinophils: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Eosinophils: change at week 2 | -0.019 (0.1087) | -0.000 (0.0734) | -0.023 (0.0809) | 0.009 (0.0980) | -0.029 (0.0915) | -0.006 (0.0621) | 0.022 (0.0762) | 0.005 (0.1256)
  Eosinophils: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Eosinophils: change at week 4 | 0.032 (0.1813) | 0.018 (0.1120) | 0.008 (0.1325) | -0.019 (0.1102) | -0.032 (0.1040) | -0.012 (0.0832) | 0.042 (0.1076) | -0.012 (0.1499)
  Eosinophils: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Eosinophils: change at week 6 | 0.002 (0.0935) | 0.029 (0.1090) | -0.025 (0.1351) | 0.018 (0.1387) | -0.027 (0.1125) | -0.007 (0.1025) | -0.001 (0.0812) | -0.022 (0.1415)
  Eosinophils: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Eosinophils: change at follow-up visit | 0.022 (0.1461) | 0.006 (0.0931) | -0.023 (0.1196) | -0.004 (0.1810) | 0.008 (0.1270) | -0.008 (0.2483) | 0.048 (0.1520) | -0.011 (0.1945)
  Monocytes: change at week 1: number analyzed (Participants) | 34 | 35 | 32 | 34 | 34 | 33 | 35 | 34
  Monocytes: change at week 1 | 0.006 (0.1796) | 0.030 (0.0855) | 0.030 (0.0987) | 0.009 (0.0879) | 0.019 (0.1055) | 0.006 (0.0877) | 0.051 (0.1244) | 0.011 (0.1195)
  Monocytes: change at week 2: number analyzed (Participants) | 34 | 33 | 32 | 34 | 32 | 30 | 33 | 31
  Monocytes: change at week 2 | -0.006 (0.1509) | 0.016 (0.1343) | -0.003 (0.0724) | -0.014 (0.1055) | 0.017 (0.0865) | 0.013 (0.0983) | 0.049 (0.1471) | 0.025 (0.1496)
  Monocytes: change at week 4: number analyzed (Participants) | 28 | 27 | 33 | 31 | 32 | 25 | 30 | 30
  Monocytes: change at week 4 | -0.035 (0.1904) | 0.030 (0.1212) | 0.013 (0.1234) | -0.003 (0.1092) | 0.009 (0.0986) | 0.035 (0.0978) | 0.007 (0.1008) | 0.038 (0.1331)
  Monocytes: change at week 6: number analyzed (Participants) | 29 | 27 | 31 | 32 | 31 | 24 | 32 | 33
  Monocytes: change at week 6 | 0.017 (0.1777) | 0.017 (0.1069) | -0.025 (0.1191) | -0.005 (0.1021) | -0.019 (0.0726) | 0.004 (0.0847) | 0.003 (0.1097) | -0.012 (0.1200)
  Monocytes: change at follow-up visit: number analyzed (Participants) | 30 | 29 | 30 | 32 | 30 | 31 | 32 | 30
  Monocytes: change at follow-up visit | 0.011 (0.1806) | 0.021 (0.0824) | 0.030 (0.1467) | 0.005 (0.0887) | 0.021 (0.0739) | 0.018 (0.1047) | 0.029 (0.1788) | -0.006 (0.1282)

20. Secondary Outcome: Change From Baseline in Lipids Profile Values at Week 6
Description: Lipid parameters that were assessed: high density lipoprotein (HDL) cholesterol, triglycerides, cholesterol, low density lipoprotein (LDL) cholesterol.
Time Frame: Baseline, Week 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Microgram per deciliter
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 28 | 27 | 31 | 32 | 29 | 24 | 30 | 32
Microgram per deciliter
  HDL cholesterol | -2.8 (6.65) | 0.1 (5.34) | -1.3 (7.74) | 2.7 (8.33) | 1.9 (11.18) | 0.0 (6.76) | 1.2 (4.12) | 0.3 (8.56)
  Triglycerides: number analyzed (Participants) | 28 | 27 | 31 | 31 | 29 | 24 | 30 | 32
  Triglycerides | 3.3 (38.84) | -4.2 (59.30) | -6.5 (37.30) | 1.8 (60.74) | -18.9 (56.78) | -8.1 (50.41) | -7.0 (58.36) | -4.4 (55.66)
  Cholesterol | -3.5 (16.39) | -5.6 (27.59) | -12.8 (20.53) | 6.8 (24.09) | -10.4 (30.79) | -0.2 (18.70) | 5.3 (30.58) | -0.9 (19.86)
  LDL Cholesterol | -3.4 (14.45) | -6.3 (25.28) | -12.1 (16.44) | 2.1 (20.13) | -11.0 (29.06) | -0.8 (14.48) | 4.4 (23.55) | -1.1 (16.29)

21. Secondary Outcome: Change From Baseline in Ratio of LDL Cholesterol to HDL Cholesterol Lipids Profile at Week 6
Description: Mean change in total cholesterol/HDL cholesterol ratio was assessed and reported.
Time Frame: Baseline, Week 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 28 | 27 | 31 | 32 | 29 | 24 | 30 | 32
Ratio | 0.0 (0.31) | -0.1 (0.48) | -0.2 (0.40) | -0.0 (0.32) | -0.3 (0.77) | -0.0 (0.35) | 0.0 (0.46) | -0.0 (0.42)

22. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter- Heart Rate at Weeks 2 and 6
Time Frame: Baseline, Weeks 2 and 6
Population: Safety analysis set included all participants who were randomly assigned to study drug and who applied at least 1 dose of study drug. Here, "number analyzed" signifies participants evaluable for the each specified time point.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Beats per minute
  Baseline | 66.8 (11.45) | 66.9 (9.33) | 68.4 (14.66) | 64.9 (9.05) | 64.9 (12.26) | 66.9 (12.03) | 68.2 (12.11) | 68.1 (12.48)
  Change at week 2: number analyzed (Participants) | 33 | 31 | 33 | 33 | 31 | 26 | 34 | 32
  Change at week 2 | 0.7 (10.05) | -0.5 (8.03) | -1.8 (11.53) | -0.6 (7.88) | 1.9 (8.01) | 2.2 (8.76) | 1.7 (9.13) | 1.7 (12.52)
  Change at week 6: number analyzed (Participants) | 28 | 27 | 33 | 32 | 30 | 24 | 31 | 33
  Change at week 6 | 0.3 (6.19) | -1.1 (7.65) | -1.7 (9.06) | 0.8 (8.53) | -0.3 (8.46) | -0.8 (8.23) | 0.5 (8.76) | -0.4 (12.06)

23. Secondary Outcome: Change From Baseline in PR, QRS, QTCF and QT Interval at Weeks 2 and 6
Time Frame: Baseline, Weeks 2 and 6
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Milliseconds
  PR interval: baseline | 161.9 (23.30) | 160.2 (24.01) | 161.4 (27.59) | 162.5 (22.04) | 160.7 (24.20) | 156.4 (22.65) | 157.9 (23.55) | 157.8 (23.15)
  PR interval: change at week 2: number analyzed (Participants) | 33 | 31 | 33 | 33 | 31 | 26 | 34 | 32
  PR interval: change at week 2 | 0.8 (14.41) | -0.9 (15.92) | 0.7 (18.54) | 0.3 (10.13) | 1.1 (14.42) | 6.0 (14.79) | 1.2 (16.06) | 2.1 (7.98)
  PR interval: change at week 6: number analyzed (Participants) | 28 | 27 | 33 | 32 | 30 | 24 | 31 | 33
  PR interval: change at week 6 | -0.9 (10.16) | -0.1 (13.81) | 2.8 (19.66) | 2.9 (13.63) | 3.5 (21.88) | 4.0 (14.56) | 6.5 (19.15) | 5.7 (16.11)
  QRS interval: baseline | 92.5 (9.36) | 91.5 (9.71) | 91.1 (9.29) | 93.0 (11.13) | 93.1 (8.69) | 92.2 (13.00) | 92.4 (13.30) | 91.5 (11.68)
  QRS interval: change at week 2: number analyzed (Participants) | 33 | 31 | 33 | 33 | 31 | 26 | 34 | 32
  QRS interval: change at week 2 | -1.4 (8.02) | -0.4 (5.34) | -1.3 (3.46) | -0.8 (5.64) | 0.1 (4.79) | 1.5 (9.29) | 0.2 (8.07) | 1.0 (5.63)
  QRS interval: change at week 6: number analyzed (Participants) | 28 | 27 | 33 | 32 | 30 | 24 | 31 | 33
  QRS interval: change at week 6 | -1.9 (6.55) | 1.4 (5.62) | -0.5 (4.76) | -0.9 (4.04) | -1.3 (4.00) | 0.9 (6.37) | 0.6 (5.49) | 0.7 (5.67)
  QTCF interval: baseline | 407.7 (17.78) | 397.9 (15.98) | 403.8 (22.43) | 408.5 (18.42) | 401.0 (16.29) | 403.0 (16.65) | 397.7 (17.05) | 405.0 (20.38)
  QTCF interval: change at week 2: number analyzed (Participants) | 33 | 31 | 36 | 33 | 31 | 26 | 34 | 32
  QTCF interval: change at week 2 | -5.7 (11.86) | -1.5 (13.70) | -3.9 (15.60) | 2.6 (16.20) | -0.6 (12.75) | 1.4 (15.56) | 2.4 (10.32) | -4.6 (15.43)
  QTCF interval: change at week 6: number analyzed (Participants) | 28 | 27 | 33 | 32 | 30 | 24 | 31 | 33
  QTCF interval: change at week 6 | -4.1 (14.61) | -0.5 (14.93) | -1.9 (14.37) | 0.3 (17.19) | -1.4 (14.93) | 4.6 (14.27) | 2.0 (11.94) | -0.2 (9.67)
  QT interval: baseline | 395.2 (31.53) | 385.3 (23.64) | 388.8 (33.66) | 401.0 (25.23) | 392.0 (27.36) | 390.9 (24.87) | 383.8 (30.79) | 390.6 (32.43)
  QT interval: change at week 2: number analyzed (Participants) | 33 | 31 | 33 | 33 | 31 | 26 | 34 | 22
  QT interval: change at week 2 | -5.9 (23.16) | -1.3 (17.73) | -1.1 (19.31) | 3.5 (21.06) | -4.5 (15.75) | 1.2 (24.03) | -2.3 (18.69) | -4.6 (25.76)
  QT interval: change at week 6: number analyzed (Participants) | 28 | 27 | 33 | 32 | 30 | 24 | 31 | 32
  QT interval: change at week 6 | -4.9 (19.54) | 1.3 (18.11) | 0.9 (16.11) | -4.1 (23.42) | -0.9 (20.12) | 7.8 (24.11) | -1.4 (20.47) | 4.0 (27.74)

24. Secondary Outcome: Change From Baseline in Vital Signs- Blood Pressure (BP) at Weeks 2 and 6
Description: Blood pressure included supine and sitting systolic and diastolic BP.
Time Frame: Baseline, Weeks 2 and 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 25 | 26 | 29 | 22 | 23 | 26 | 23 | 25
Millimeters of mercury
  Supine systolic BP: Baseline | 123.3 (12.01) | 123.2 (12.35) | 123.0 (13.89) | 119.7 (9.08) | 122.6 (12.76) | 123.1 (12.40) | 117.1 (14.07) | 118.9 (12.43)
  Supine systolic BP: change at week 2: number analyzed (Participants) | 21 | 20 | 25 | 18 | 20 | 18 | 21 | 22
  Supine systolic BP: change at week 2 | 0.3 (11.55) | -1.4 (9.61) | 0.5 (14.73) | 2.3 (6.99) | -0.3 (10.25) | -0.3 (8.02) | 3.5 (13.65) | 2.9 (8.48)
  Supine systolic BP: change at week 6: number analyzed (Participants) | 16 | 15 | 24 | 17 | 19 | 18 | 21 | 22
  Supine systolic BP: change at week 6 | -0.2 (12.98) | 1.1 (10.06) | 2.0 (14.05) | 0.2 (9.13) | -3.4 (11.02) | -1.4 (10.49) | 2.1 (12.41) | 0.6 (10.31)
  Sitting systolic BP: Baseline: number analyzed (Participants) | 15 | 17 | 17 | 19 | 19 | 16 | 18 | 15
  Sitting systolic BP: Baseline | 117.7 (13.05) | 120.8 (10.26) | 120.2 (12.43) | 116.9 (17.76) | 124.6 (11.25) | 119.4 (12.96) | 122.9 (15.25) | 125.6 (12.21)
  Sitting systolic BP: change at week 2: number analyzed (Participants) | 12 | 11 | 8 | 15 | 11 | 7 | 11 | 10
  Sitting systolic BP: change at week 2 | 1.3 (12.12) | -1.9 (11.86) | -3.9 (14.54) | 1.3 (13.59) | -2.4 (11.76) | -3.1 (10.46) | 1.1 (9.81) | 4.4 (11.68)
  Sitting systolic BP: change at week 6: number analyzed (Participants) | 12 | 10 | 9 | 15 | 10 | 5 | 10 | 11
  Sitting systolic BP: change at week 6 | 0.6 (12.24) | -7.5 (8.67) | -9.4 (8.95) | 1.0 (14.63) | -8.4 (10.81) | -0.6 (14.40) | -3.6 (8.37) | -1.5 (5.80)
  Supine diastolic BP: Baseline | 77.7 (9.28) | 75.2 (8.79) | 78.8 (8.39) | 74.5 (8.26) | 75.9 (8.78) | 77.5 (8.71) | 74.4 (8.20) | 73.7 (8.59)
  Supine diastolic BP: change at week 2: number analyzed (Participants) | 21 | 20 | 25 | 18 | 20 | 18 | 21 | 22
  Supine diastolic BP: change at week 2 | 0.5 (7.51) | 0.6 (6.47) | -0.4 (8.50) | 1.6 (10.33) | 1.2 (8.32) | -2.8 (6.69) | 1.6 (8.89) | 1.4 (7.74)
  Supine diastolic BP: change at week 6: number analyzed (Participants) | 16 | 15 | 24 | 17 | 19 | 18 | 21 | 22
  Supine diastolic BP: change at week 6 | -2.5 (7.69) | 1.5 (7.61) | -0.7 (8.32) | 0.5 (7.96) | -0.9 (10.65) | -1.6 (6.22) | 1.9 (9.72) | 0.5 (6.32)
  Sitting diastolic BP: Baseline: number analyzed (Participants) | 15 | 17 | 17 | 19 | 19 | 16 | 18 | 15
  Sitting diastolic BP: Baseline | 76.5 (9.28) | 80.1 (6.76) | 77.8 (10.02) | 69.6 (11.48) | 80.9 (8.21) | 75.1 (5.77) | 77.1 (12.00) | 80.3 (7.83)
  Sitting diastolic BP: change at week 2: number analyzed (Participants) | 12 | 11 | 8 | 15 | 11 | 7 | 11 | 10
  Sitting diastolic BP: change at week 2 | -1.6 (8.49) | 0.7 (7.93) | 0.0 (9.44) | 1.6 (12.00) | -2.9 (10.77) | 1.7 (8.20) | 4.5 (5.80) | -1.2 (6.49)
  Sitting diastolic BP: change at week 6: number analyzed (Participants) | 12 | 10 | 9 | 15 | 10 | 5 | 10 | 11
  Sitting diastolic BP: change at week 6 | 0.8 (9.90) | 0.0 (5.79) | -1.6 (11.97) | 1.1 (15.61) | -5.3 (9.27) | -2.8 (12.60) | -0.3 (7.89) | 0.4 (8.41)

25. Secondary Outcome: Change From Baseline in Vital Signs- Pulse Rate at Weeks 2 and 6
Time Frame: Baseline, Weeks 2 and 6
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Beats per minute
  Baseline | 69.6 (12.58) | 69.5 (9.82) | 72.9 (14.30) | 67.9 (9.31) | 68.8 (11.76) | 69.4 (11.15) | 70.1 (11.18) | 68.2 (9.59)
  Change at week 2: number analyzed (Participants) | 33 | 31 | 33 | 33 | 31 | 26 | 33 | 32
  Change at week 2 | 0.5 (10.41) | 0.2 (8.11) | -2.5 (9.66) | 1.1 (9.13) | 0.5 (6.54) | 3.7 (9.47) | 2.8 (8.28) | 4.1 (9.16)
  Change at week 6: number analyzed (Participants) | 28 | 27 | 33 | 32 | 30 | 24 | 31 | 33
  Change at week 6 | 2.1 (10.59) | 0.3 (8.04) | -1.4 (11.90) | 0.9 (9.71) | 1.8 (8.73) | 4.1 (6.76) | 0.5 (9.12) | 1.8 (8.64)

26. Secondary Outcome: Change From Baseline in Vital Signs- Temperature at Weeks 2 and 6
Time Frame: Baseline, Weeks 2 and 6
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Degree Celsius
  Baseline | 36.5 (0.33) | 36.5 (0.43) | 36.6 (0.44) | 36.6 (0.33) | 36.5 (0.37) | 36.5 (0.29) | 36.6 (0.41) | 36.6 (0.29)
  Change at week 2: number analyzed (Participants) | 33 | 31 | 33 | 33 | 31 | 26 | 33 | 32
  Change at week 2 | -0.1 (0.41) | -0.1 (0.30) | 0.0 (0.38) | -0.0 (0.43) | 0.1 (0.35) | -0.0 (0.38) | 0.0 (0.34) | 0.0 (0.41)
  Change at week 6: number analyzed (Participants) | 28 | 27 | 33 | 32 | 30 | 24 | 31 | 33
  Change at week 6 | -0.0 (0.40) | -0.0 (0.29) | 0.0 (0.38) | 0.1 (0.32) | 0.0 (0.29) | 0.1 (0.50) | 0.0 (0.37) | -0.0 (0.46)

27. Secondary Outcome: Number of Participants With Each Severity Grade in Local Tolerability Assessments
Description: Local tolerability skin assessments were performed by the investigator and graded based on severity from grade 0 to 4 as: grade 0=none (no evidence of local intolerance); grade 1=mild (minimal erythema and/or oedema, slight glazed appearance); grade 2= moderate (definite erythema and/or oedema with peeling and/or cracking but needs no adaptation of posology) grade 3=severe (erythema, oedema glazing with fissures, few vesicles or papules consider removing topical agent [if still in place]) and grade 4= very severe (strong reaction spreading beyond the treated area, bullous reaction, erosions: removal of topical agent [if still in place]). Higher grades indicated worsening of condition. Only those categories in which at least 1 participant had data were reported.
Time Frame: Day 1 and any day on of Week 1, 2, 4, 6: pre dose (before application of IP) and post dose (after application of IP); Follow up visit (28 days after last dose of study drug = maximum up to Day 71) and Early termination (anytime within week 11)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
Number analyzed (Participants) | 37 | 37 | 36 | 37 | 36 | 36 | 36 | 37
Participants
  Day 1: tolerability before: none | 35 | 35 | 31 | 33 | 36 | 35 | 34 | 36
  Day 1: tolerability before: mild | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 0
  Day 1: tolerability before: moderate | 2 | 2 | 4 | 1 | 0 | 0 | 0 | 1
  Day 1: tolerability after: none | 33 | 36 | 30 | 33 | 35 | 34 | 32 | 33
  Day 1: tolerability after: mild | 1 | 0 | 1 | 2 | 0 | 2 | 4 | 1
  Day 1: tolerability after: moderate | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
  Week 1: tolerability before: none | 31 | 28 | 28 | 30 | 30 | 30 | 33 | 33
  Week 1: tolerability before: mild | 1 | 2 | 3 | 3 | 3 | 1 | 1 | 1
  Week 1: tolerability before: moderate | 2 | 0 | 3 | 0 | 0 | 1 | 0 | 0
  Week 1: tolerability after: none | 28 | 29 | 29 | 30 | 28 | 27 | 32 | 31
  Week 1: tolerability after: mild | 2 | 2 | 2 | 3 | 2 | 3 | 1 | 1
  Week 1: tolerability after: moderate | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0
  Week 2: tolerability before: none | 29 | 28 | 26 | 30 | 30 | 23 | 31 | 33
  Week 2: tolerability before: mild | 3 | 2 | 2 | 2 | 1 | 1 | 0 | 0
  Week 2: tolerability before: moderate | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0
  Week 2: tolerability after: none | 28 | 26 | 29 | 31 | 29 | 23 | 32 | 30
  Week 2: tolerability after: mild | 1 | 3 | 2 | 1 | 1 | 2 | 0 | 1
  Week 2: tolerability after: moderate | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
  Week 4: tolerability before: none | 27 | 26 | 30 | 30 | 30 | 24 | 31 | 31
  Week 4: tolerability before: mild | 0 | 2 | 2 | 2 | 0 | 0 | 1 | 1
  Week 4: tolerability before: moderate | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
  Week 4: tolerability after: none | 24 | 26 | 30 | 30 | 29 | 24 | 31 | 30
  Week 4: tolerability after: mild | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 0
  Week 4: tolerability after: moderate | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Week 6: tolerability before: none | 26 | 25 | 29 | 30 | 30 | 21 | 30 | 32
  Week 6: tolerability before: mild | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1
  Week 6: tolerability before: moderate | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
  Week 6: tolerability after: none | 25 | 24 | 28 | 29 | 29 | 22 | 30 | 30
  Week 6: tolerability after: mild | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
  Week 6: tolerability after: moderate | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  Early termination:tolerability: none | 6 | 5 | 3 | 2 | 2 | 9 | 2 | 1
  Early termination:tolerability: mild | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  Early termination:tolerability: moderate | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Early termination:tolerability: severe | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Follow Up: tolerability: none | 22 | 26 | 25 | 25 | 28 | 25 | 26 | 28
  Follow Up: tolerability: mild | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1
  Follow Up: tolerability: moderate | 1 | 0 | 1 | 4 | 1 | 1 | 0 | 0
  Follow Up: tolerability: severe | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to at least 28 days after last dose of study drug (approximately up to Week 11)
Arm/Group | Vehicle Cream Once Daily (QD) | PF-06700841 0.1% Cream QD | PF-06700841 0.3% Cream QD | PF-06700841 1.0% Cream QD | PF-06700841 3.0% Cream QD | Vehicle Cream Twice Daily (BID) | PF-06700841 0.3% Cream BID | PF-06700841 1.0% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/36 | 0/37 | 0/36 | 0/36 | 0/36 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/36 | 0/37 | 0/36 | 0/36 | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 18/37 | 17/37 | 11/36 | 12/37 | 10/36 | 17/36 | 9/36 | 14/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Cream Once Daily (QD) (N=37) | PF-06700841 0.1% Cream QD (N=37) | PF-06700841 0.3% Cream QD (N=36) | PF-06700841 1.0% Cream QD (N=37) | PF-06700841 3.0% Cream QD (N=36) | Vehicle Cream Twice Daily (BID) (N=36) | PF-06700841 0.3% Cream BID (N=36) | PF-06700841 1.0% Cream BID (N=37)
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Administration site warmth (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site acne (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Application site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Application site pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Application site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cockroach allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mite allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial allergy (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Kaposi's varicelliform eruption (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 3 | 4 | 2 | 2 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipids abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 0 | 1 | 3 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Solar urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT03903822/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03903822/SAP_001.pdf